| <b>Document Type:</b> | Study Protocol |
|---|---|
| Official Title: | A multicenter, randomized, placebo-controlled, parallel group, double blind, dose-finding Phase II trial to study the efficacy, safety, pharmacokinetic and pharmacodynamic effects of the oral partial adenosine A1 receptor agonist neladenoson bialanate over 20 weeks in patients with chronic heart failure with reduced ejection fraction |
| NCT Number: | NCT02992288 |
| <b>Document Date:</b> | 17 FEB 2017 |



17 FEB 2017 Version: 2.0 

# Cover page of the integrated protocol

A multicenter, randomized, placebo-controlled, parallel group, double blind, dose-finding Phase II trial to study the efficacy, safety, pharmacokinetic and pharmacodynamic effects of the oral partial adenosine A1 receptor agonist neladenoson bialanate over 20 weeks in patients with chronic heart failure with reduced ejection fraction

This protocol version is an integration of the following documents / sections:

- Original protocol, Version 1.0, dated 31 OCT 2016
- Amendment no. 2 (described in Section 15.1) forming integrated protocol Version 2.0, dated 17 FEB 2017

Amendments not included in the consecutive numbering of amendments are local amendments not forming part of this integrated global protocol.




# 1. Title page

A multicenter, randomized, placebo-controlled, parallel group, double blind, dose-finding Phase II trial to study the efficacy, safety, pharmacokinetic and pharmacodynamic effects of the oral partial adenosine A1 receptor agonist neladenoson bialanate over 20 weeks in patients with chronic heart failure with reduced ejection fraction

Short title: PANTHEON

Test drug: neladenoson bialanate / BAY 1067197

Study purpose: dose finding

Clinical study phase: IIb Date: 17 FEB 2016

Registration: EudraCT no.: 2016-003839-38 Version no.: 2.0

Sponsor's study no.: BAY 1067197 / 15128

Sponsor: Non-US: Bayer AG, D-51368 Leverkusen, Germany

US territory: Bayer HealthCare Pharmaceuticals Inc., 100 Bayer Boulevard, P.O. Box 915, Whippany NJ 07981-0915, USA

Sponsor's medical

expert:

PPD PPD

Bayer Vital GmbH

Kaiser-Wilhelm-Allee 70 / K56 51368, Leverkusen, Germany

Phone: PPD Email: PPD

The study will be conducted in compliance with the protocol, ICH-GCP and any applicable regulatory requirements.

#### Confidential

The information provided in this document is strictly confidential and is intended solely for the guidance of the clinical investigation. Reproduction or disclosure of this document - whether in part or in full - to parties not associated with the clinical investigation, or its use for any other purpose, without the prior written consent of the sponsor is not permitted.

Throughout this document, symbols indicating proprietary names (®, TM) may not be displayed. Hence, the appearance of product names without these symbols does not imply that these names are not protected.



17 FEB 2017

Version: 2.0


# Signature of the sponsor's medically responsible person

The signatory agrees to the content of the final integrated clinical study protocol as presented.

Name: PPD Role: Global Clinical Leader

PPD

Date: 17/2/2017 Signature:




# Signature of principal investigator

| The signatory agrees to the content of the final c | clinical study protocol as presented. |
|---|---|
| Name: | |
| Affiliation: | |
| Date: Si | ignature: |
| Signed copies of this signature page are stored in center's investigator site file. | n the sponsor's study file and in the respective |




# 2. Synopsis

| Title | A multicenter, randomized, placebo-controlled, parallel group, double blind, dose-finding Phase II trial to study the efficacy, safety, pharmacokinetic and pharmacodynamic effects of the oral partial adenosine A1 receptor agonist neladenoson bialanate over 20 weeks in patients with chronic heart failure with reduced ejection fraction |
|---|---|
| Short title | PANTHEON |
| Clinical study phase | IIb |
| Study objective(s) | The objective of the study is to find the optimal dose of neladenoson bialanate for the Phase III trial by detecting and characterizing a significant doseresponse relationship in the two primary efficacy endpoints, absolute change from baseline in left ventricular ejection fraction (LVEF) and log-transformed NT-proBNP at 20 weeks, in patients with chronic heart failure with reduced ejection fraction (HFrEF), and by characterizing the safety, tolerability and pharmacodynamic effects of the compound when given in addition to standard therapy for HFrEF. |
| | An exploratory objective is to further assess pharmacokinetic parameters and blood and urine biomarkers. |
| Test drug(s) | |
| Name of active ingredient | neladenoson bialanate |
| Dose(s) | 5 mg, 10 mg, 20 mg, 30 mg, and 40 mg once daily |
| Route of administration | Oral |
| <b>Duration of treatment</b> | 20 weeks |
| Reference drug(s) | |
| Name of active ingredient | Placebo |
| Dose(s) | Not applicable |
| Route of administration | Oral |
| <b>Duration of treatment</b> | 20 weeks |
| Background treatment | Standard therapy for heart failure given concomitantly with the test drug / placebo |
| Indication | Chronic heart failure (NYHA class II-IV) with reduced ejection fraction |
| Diagnosis and main criteria for inclusion | <ol> <li>Men or women aged 18 years and older</li> <li>Diagnosis of chronic heart failure, NYHA class II-IV, LVEF ≤ 35% assessed by any imaging modality (e.g. echocardiography, cardiac magnetic resonance, cine levocardiography) within 6 months prior to runin: if several values are available the last assessment of LVEF should be ≤ 35%.</li> </ol> |
| | <ul> <li>3. One of the following (or both),</li> <li>a) Worsening chronic heart failure requiring hospitalization or an unscheduled outpatient visit in the last 3 months, both requiring initiation or intensification of heart failure therapy and with either:</li> <li>○ BNP ≥ 100 pg/mL or NT-proBNP ≥400 pg/mL (sinus rhythm) or</li> <li>○ BNP ≥ 300 pg/mL or NT-proBNP ≥1200 pg/mL (atrial fibrillation)</li> </ul> |




| AND/OR |
|--------|

#### b) at any time in the past 4 weeks one of:

- o BNP  $\geq$  300 pg/mL or NT-proBNP  $\geq$  1200 pg/mL (sinus rhythm)
- $\circ \quad BNP \geq 600 \; pg/mL \; or \; NT\text{-pro}BNP \geq 2400 \; pg/mL \; (atrial \; fibrillation)$

For patients on treatment with angiotensin receptor-neprilysin inhibitors (ARNIs), e.g. Entresto only NT-proBNP values can be used to assess eligibility.

4. Written informed consent before any study-specific procedure

# Diagnosis and main criteria for exclusion

- 1. Acute de-novo heart failure
- 2. Requirement of any of the following 48 hours prior to randomization:
  - o Intravenous (IV) vasodilating drugs (e.g. nitrates, nitroprusside)
  - IV natriuretic peptides (e.g. nesiritide, carperitide)
  - IV positive inotropic agents
  - o IV diuretics
  - o IV antibiotics
  - Mechanical support (e.g. intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device)
- 3. Any cause of chronic heart failure other than ischemic cardiomyopathy and idiopathic dilated cardiomyopathy
- 4. Known clinically significant persistent coronary ischemia based on medical history, preexisting or current exercise testing
- 5. Occurrence of any of the following within 3 months prior to randomization:
  - o Myocardial infarction
  - o Hospitalization for unstable angina
  - o Stroke or transient ischemic attack
  - o Coronary artery bypass graft (CABG)
  - o Percutaneous coronary intervention (PCI)
  - o Implantation of a cardiac resynchronization therapy device (CRTD)
  - o Carotid angioplasty
- 6. PCI, CABG or implantation of a CRTD planned between randomization and end of study
- 7. Sustained \* systolic blood pressure ≤ 90 mmHg and / or signs and symptoms of hypotension prior to randomization
- 8. Sustained \* systolic blood pressure ≥ 160 mmHg
- 9. Sustained \* bradycardia with heart rate < 50 beats/minute or tachycardia with heart rate > 100 beats/minute prior to randomization
- Known clinically relevant ventricular arrhythmias (sustained ventricular tachycardia, ventricular flutter or fibrillation) within 3 months prior to consent based on either medical history or implantable cardioverter defibrillator (ICD)-testing results (if applicable)
- 11. Clinically relevant permanent or intermittent atrioventricular (AV)-block  $\geq$  grade II in patients without a permanent pacemaker or ICD / CRTD
- 12. Severe valvular disease with indicated or planned valve repair / replacement
- 13. Listing for heart transplantation and / or anticipated implantation of a ventricular assist device




- 14. Severe pulmonary disease with any of the following:
  - o Requirement of continuous (home) oxygen or
  - o History of chronic obstructive pulmonary disease ≥ GOLD III or
  - o Use of systemic corticosteroids
- 15. Asthma bronchiale with any of the following:
  - o Symptoms not well-controlled within the past 6 months or
  - o Ever intubated or in an intensive care unit for asthma
- 16. Anemia with hemoglobin < 10 g/dL within 3 months prior to randomization. If several values are available the latest result should be used
- 17. Body mass index (BMI) > 40 kg/m<sup>2</sup> at randomization or a history of poor quality LVEF measurement by echocardiography
- 18. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m<sup>2</sup> calculated by Modification of Diet in Renal Disease (MDRD) formula within 3 months prior to randomization. If several values are available the latest result should be used.
- 19. Hepatic insufficiency classified as Child-Pugh B or C, or any of the following:
  - o Primary biliary cirrhosis (PBC)
  - o Primary sclerosing cholangitis
  - o PBC-autoimmune hepatitis overlap syndrome
- 20. Concomitant use of any of the following therapy that cannot be discontinued:
  - Moderate or strong CYP3A4 inhibitors (Of note: grapefruit is a strong CYP3A4 inhibitor.)
  - o CYP3A4 inducers
  - Strong CYP2C8 inhibitors (Of note: clopidogrel is a strong CYP2C8 inhibitor)
  - Theophylline
  - Drugs having significant pre-systemic clearance via UGT1A1 in the intestine

Respective substances must be stopped at least 7 days before randomization.

- 21. Women of childbearing potential (women are considered of childbearing potential if they are not surgically sterile or postmenopausal, defined as amenorrhea for > 12 months)
- 22. Any condition or therapy, which would make the patient unsuitable for the study, or life expectancy less than 12 months (e.g. active malignancy)
- 23. Known current heavy alcohol consumption or the use of illicit drugs that, in the opinion of the investigator, may interfere with the patient's safety and / or compliance
- 24. Previous (within 30 days or 5 half-lives of the investigational drug, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s)
- 25. Previous assignment to treatment during this study
- 26. Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site)



| | No. BAY 106/19// 15128 | R |
|---|---|---|
| | 27. Known allergies, intolerance or hypersensitivities to the stu (active substance or excipients), adhesives or hydrogel | dy treatment |
| | * At two consecutive visits | |
| Study design | Randomized, double-blind, placebo-controlled, parallel-group, r | nulticenter |
| Methodology | The study will comprise a 1-week run-in period, 20-week treatm a 6-week follow-up period (27 weeks total). | • |
| | Patients will have site visits at weeks -1, 0 (baseline), 4, 8, 12, 2 treatment visit) and 24 (safety follow-up visit). In addition, 2 ph weeks 2 and 26 will be made to assess patients' safety, and one phone call - to remind the patients of AVIVO self-application at | one calls at additional |
| | LVEF will be measured by echocardiography at baseline and en NT-proBNP will be measured at baseline, Week 4 and end of travill be monitored throughout the study. PK samples will be taked patients at dedicated time points. Additional biomarkers reflecting pharmacodynamic activity of the drug will be examined, as well biomarkers that may predict drug response. | eatment. Safety<br>en from all<br>ng the |
| Type of control | Placebo control | |
| <b>Data Monitoring Committee</b> | Yes | |
| Number of patients | Approximately 384 patients are planned to be randomized. | |
| Primary variables | • Absolute change from baseline in left ventricular ejection frac<br>%) after 20 weeks of treatment measured by echocardiograph | |
| | <ul> <li>Absolute change from baseline in log-transformed NT-proBN<br/>after 20 weeks, i.e., log-transformed NT-proBNP at Week 20<br/>transformed NT-proBNP at baseline.</li> </ul> | |
| Time point / frame of<br>measurement for<br>primary variables | After 20 weeks of treatment | |
| Plan for statistical analysis | The primary efficacy analysis will be performed on the primary variables in patients belonging to the per-protocol set using a typ 5%. | |
| | For the assessment of a dose-response relationship in the change NT-proBNP, the MCP-Mod method, combining multiple compa procedures (MCP) principles with modeling techniques under muncertainty, will be used. | arison |
| | The overall outcome of the primary efficacy analysis will be conpositive if at least one of the two null hypotheses related to the parailles can be rejected. The Hochberg (step-up) procedure will control the family-wise error rate. | orimary efficacy |
| | A set with 5 candidate dose-response models has been specified detection of a dose-response signal, each of the dose-response meandidate set will be tested at the corresponding type I error level sided multiple contrast test based on pre-specified contrast coeff dose-response signal is established, a dose-response model will data and target dose(s) of interest will be estimated based on the dose-response model. Other efficacy variables will be analyzed analogously to the prinor descriptively. | nodels in the el, using a one-<br>ficients. If a be fitted to the estimated |




# **Table of contents**

| Cov | ver page of the integrated protocol | 1 |
|------------|--------------------------------------------------------|----|
| 1. | Title page | 2 |
| 2. | Synopsis | 5 |
| Tab | ole of contents | 9 |
| | ole of tables | |
| | ole of figures | |
| List | t of abbreviations | 12 |
| 3. | Introduction | |
| 3.1 | Background | |
| 3.2<br>3.3 | Partial adenosine A1 receptor agonism in heart failure | |
| 3.4 | Rationale of the study | |
| <b>4.</b> | Study objectives | |
| 5. | Study design | |
| 5.1 | Design overview | |
| 5.2 | Primary variables | |
| 5.3 | Justification of the design | |
| 5.4 | End of study | |
| 6. | Study population | 21 |
| 6.1 | Inclusion criteria | |
| 6.2 | Exclusion criteria | 22 |
| 6.3 | Justification of selection criteria | 24 |
| 6.4 | Withdrawal of patients from study | 24 |
| 6.4. | 1 Withdrawal | 24 |
| 6.4. | 1 | |
| 6.5 | Patient identification | 26 |
| <b>7.</b> | Treatments | |
| 7.1 | | |
| 7.2 | Identity of study treatment | |
| 7.3 | Treatment assignment | |
| 7.4 | Dosage and administration. | |
| 7.5 | Blinding | |
| 7.6 | Drug logistics and accountability | |
| 7.7 | Treatment compliance | 29 |
| 8. | Non-study therapy | |
| 8.1 | Prior and concomitant therapy | |
| 8.1. | | |
| 8.1. | 1 3 | |
| 8.2 | Post-study therapy | 31 |




| 9. Procedures and variables | 31 |
|---|---|
| 9.1 Tabular schedule of evaluations | 31 |
| 9.2 Visit description | 34 |
| 9.2.1 Visit 1 (Week -1, run-in) | 34 |
| 9.2.2 Visit 2 (Week 0, baseline) | 34 |
| 9.2.3 Visit 3 (Week 2, phone call) | 35 |
| 9.2.4 Visit 4 (Week 4) | 35 |
| 9.2.5 Visit 5 (Week 8) | 36 |
| 9.2.6 Visit 6 (Week 12) | 36 |
| 9.2.7 Reminder phone call at Week 19 | 37 |
| 9.2.8 Visit 7 (Week 20, EOT or premature discontinuation) | 37 |
| 9.2.9 Visit 8 (Week 24, safety follow-up) | |
| 9.2.10 Visit 9 (Week 26, phone call) | 38 |
| 9.2.11 Unscheduled Visit | 38 |
| 9.3 Population characteristics | |
| 9.3.1 Demographic and vital signs | 39 |
| 9.3.2 Medical history | |
| 9.3.3 Other baseline characteristics | |
| 9.4 Efficacy. | |
| 9.4.1 Echocardiography | |
| 9.4.2 Biomarker investigations | |
| 9.4.3 Clinical efficacy variables | |
| 9.4.4 Patient-reported outcomes | |
| 9.5 Pharmacokinetics / pharmacodynamics | |
| 9.6 Safety | |
| 9.6.1 Adverse events | |
| 9.6.2 Pregnancies | 50 |
| 9.6.3 Further safety. | |
| 9.7 Other procedures and variables. | |
| 9.8 Appropriateness of procedures / measurements | |
| 10. Statistical methods and determination of sample size | |
| 10.1 General considerations | |
| 10.2 Analysis sets | |
| 10.3 Variables and planned statistical analyses | |
| 10.3.1 Variables | |
| 10.3.2 Statistical and analytical plans. | |
| 10.3.2 Statistical and analytical plans | |
| 10.4 Determination of sample size | |
| 10.5 Planned interim analyses | |
| , and the second se | |
| 11. Data handling and quality assurance | |
| 11.1 Data recording. | |
| 11.2 Monitoring | |
| 11.3 Data processing | |
| 11.4 Missing data | |
| 11.5 Audit and inspection | 68 |




| | 1 480. 11 01 07 |
|---|---|
| 11.6 Archiving | 68 |
| 12. Premature termination of the study | 69 |
| 13. Ethical and legal aspects | 69 |
| 13.1 Investigator(s) and other study personnel | 69 |
| 13.2 Funding and financial disclosure | 71 |
| 13.3 Ethical and legal conduct of the study | |
| 13.4 Patient information and consent | |
| 13.5 Publication policy and use of data | |
| 13.6 Compensation for health damage of patients / insurance | |
| 13.7 Confidentiality | |
| 14. Reference list | |
| 15. Protocol amendments | |
| 15.1 Amendment 2 | |
| 15.1.1 Overview of changes | |
| 15.1.2 Changes to the protocol text | |
| 16. Appendices | 87 |
| 16.1 Calculating glomerular filtration rate | |
| 16.2 Calculating the Child-Pugh score | 87 |
| Table of tables | |
| Table 7–1: Identity of neladenoson bialanate (BAY 1067197) | 27 |
| Table 7–2: Identity of placebo | |
| Table 7–3: Assignment of tablets to dose groups | |
| Table 9–1: Schedule of evaluations | 32 |
| Table 9–2: Sample types used for biomarker investigations | |
| Table 9–3: Liver function monitoring | |
| Table 10–1: Dose-response shapes used in the candidate set | 58 |
| Table 10-2: Power for multiple contrast test for set of different a | ternatives |
| Table 16–1: Grading of severity of liver disease | |
| Table 16–2: Classification using the added score from Table 16– | 1 87 |
| Table of figures | |
| <b>o</b> | 20 |
| Figure 5–1: Study design overview. | |
| Figure 9–1: KCCQ Scores | |
| rigure 10–1. Dose-response snapes used in the candidate set for ( | mange in L v EF 39 |




# List of abbreviations

A1R A1 receptor

ACE angiotensin-converting enzyme

ACEi ACE inhibitor

ADHF acute decompensated heart failure

ADP adenosine diphosphate

AE(s) adverse event(s)
AF atrial fibrillation

ALT alanine aminotransferase AP alkaline phosphatase

ARB(s) angiotensin receptor blocker(s)

ARNI(s) angiotensin receptor-neprilysin inhibitor(s)

AST aspartate aminotransferase ATP adenosine triphosphate

AUC area under the time-concentration curve

AV atrioventricular

BCRP breast cancer resistance protein

BMI body mass index

BNP b-type natriuretic peptide

BSA body surface area

CABG coronary artery bypass graft cAD coronary artery disease

CE mark European Conformity mark (Conformité Européenne)

CEC Clinical Events Committee

CHF chronic heart failure

CI cardiac index CK creatine kinase

CKD chronic kidney disease

C<sub>max</sub> maximum drug concentration in plasma

CO cardiac output CRF case report form

CRO contract research organization

CRTD cardiac resynchronization therapy device

CV cardiovascular CYP cytochrome P450

DBP diastolic blood pressure
DMC Data Monitoring Committee
e.g. for example (exempli gratia)

EC(s) Ethics Committee(s)




ECG electrocardiogram eCRF electronic CRF

EDC electronic data capture

EF ejection fraction

eGFR estimated glomerular filtration rate

EOT end of treatment

EQ-5D-5L EuroQol Group 5-dimensional, 5-level questionnaire

ESC European Society of Cardiology

EU European Union

EWDT E-wave deceleration time

FAS full analysis set

FDA (US) Food and Drug Administration

FFA free fatty acids
FU follow up
g gram
Gal-3 galectin-3

GCP Good Clinical Practice

GDF-15 growth differentiation factor 15

GFR glomerular filtration rate

GGT gamma glutamyl transpeptidase GMP Good Manufacturing Practice

GOLD Global Initiative for Chronic Obstructive Lung Disease

HbA1c hemoglobin A1c HCl hydrochloride

HDL high-density lipoprotein

HF heart failure

HFpEF heart failure with preserved ejection fraction HFrEF heart failure with reduced ejection fraction

HR heart rate

hs-TNT high sensitivity troponin T

i.e. that is (*id est*)

IB investigator's brochure

ICD implantable cardioverter defibrillator

ICF informed consent form

ICH International Conference on Harmonization

IDMS Isotope dilution mass spectroscopy
IEC Independent Ethics Committee
INR international normalized ratio
IRB Institutional Review Board

ITT intent-to-treat




IV intravenous(ly)

IVSD interventricular septum diameter

IxRS interactive web / voice response system KCCQ Kansas City cardiomyopathy questionnaire

LA left atrial LAV LA volume

LAVI LA volume index
LDH lactate dehydrogenase
LDL low-density lipoprotein

LV left ventricular

LVEDV LV end-diastolic volume

LVEDVI LVEDV index

LVEF left ventricular ejection fraction LVESV left ventricular end-systolic volume

LVESVI LVESV index

MAP mean arterial pressure

MCH mean corpuscular hemoglobin

MCHC MCH concentration

MCP multiple comparison procedures

MCV mean corpuscular volume

MDRD modification of diet in renal disease

MedDRA Medical Dictionary for Regulatory Activities

mg milligram
min minute
mL milliliter

mmHg millimeter of mercury

MR-proANP mid-regional pro-atrial natriuretic peptide MRA mineralocorticoid receptor antagonist NGAL neutrophil gelatinase-associated lipocalin

NONMEM non-linear mixed effect modeling

NT-proBNP N-terminal pro-hormone b-type natriuretic peptide

NYHA New York Heart Association

OPN osteopontin

PASP pulmonary artery systolic pressure

PBC primary biliary cirrhosis

PCI percutaneous coronary intervention

PD pharmacodynamic

PDV premature discontinuation visit

Pes end-systolic pressure

pg picogram




PK pharmacokinetic PKS PK analysis set PP pulse pressure PPS per-protocol set

PTT partial thromboplastin time PWT posterior wall thickness

QC quality control

QTcB QT interval frequency-corrected according to Bazett's formula

RV right ventricular

SAC systemic arterial compliance SAE(s) serious adverse event(s) SAF safety analysis set SAP statistical analysis plan SBP systolic blood pressure

SERCA sarcoplasmic reticulum calcium adenoside triphosphatase

sST2 soluble suppression of tumorigenicity-2

SUSAR(s) suspected unexpected serious adverse reaction(s)

SV stroke volume SVI SV index

SVT(s) supraventricular tachycardia(s)

TAPSE tricuspid annular plane systolic excursion

TD tissue Doppler

TIMP-4 tissue inhibitor of metalloproteinase-4

TPR total peripheral resistance

UACR urine albumin-to-creatinine ratio

UGT1A1 uridine diphosphate glucuronosyltransferase 1A1

ULN upper limit of normal

US, USA United States (of America) VAS visual analogue scale

WCHF worsening chronic heart failure




#### 3. Introduction

# 3.1 Background

Chronic heart failure (CHF) is a major public health problem characterized by significant mortality, frequent hospitalizations, and poor quality of life, with an overall prevalence that is increasing throughout the world. The European Society of Cardiology (ESC) represents countries with a population of > 900 million, and there are at least 15 million patients with heart failure (HF) in those 51 countries (1). An estimated 5.7 million patients have HF in the United States (US) with increasing prevalence, and the incidence approaches 10 per 1000 population after 65 years of age; the lifetime risk for developing HF is one in five for men and women (2). In developed countries 1–2% of the adult population has HF, with the prevalence rising to  $\geq$  10% among persons 80 years of age or older (3). HF carries a prognosis comparable to many forms of cancer with a 5-year survival rate of approximately 50% (4), which exceeds that of many cancers (5).

Frequent hospitalizations, along with other direct and indirect costs, also place an enormous financial burden on healthcare systems; more is spent annually in the US for the treatment of HF by Medicare than on any other Medicare-covered condition (6).

The pathophysiology and clinical constellation of patients hospitalized for HF differ substantially from ambulatory patients with HF. Each episode of acute hospitalization for HF occurring annually in up to 30% of HF patients with NYHA class III and IV indicates an unfavorable underlying pathophysiology and prognosis within the course of HF (7). These patients represent an important subpopulation of patients with HF, which is denominated as worsening CHF (WCHF).

The current treatment paradigm for patients with HF with reduced ejection fraction (HFrEF) centers on systemic blockade of the maladaptive neurohumoral response, notably the enhanced and sustained activities of the sympathetic and renin-angiotensin-aldosterone systems, with hemodynamically active medications that decrease cardiac workload by reducing heart rate, preload and afterload (8-10). For patients with stable chronic HFrEF neurohumoral antagonists such as ACE inhibitors, angiotensin receptor, aldosterone and beta-blockers improve prognosis and are standard of care therapies. However, upon hospitalization for HFrEF mortality and re-hospitalization for HF remain high despite treatment with these neurohumoral blockers, indicating that this does not fully explore the complexity of HF pathophysiology.

Additionally, the repeated stepwise addition of hemodynamically active medications raises tolerability and safety concerns (e.g. hypotension and bradycardia) (11). Likewise, the high failure rate of Phase III HFrEF trials in recent years suggests that incremental benefit using the current approach may be difficult or unattainable (12), and hemodynamic compromise represents a frequent reason for failed HF drug development (13).

Therefore, addressing the failing heart directly and getting viable but not functional myocardium back to work might be a new option for the development of the next generation of hemodynamically silent HF drugs. In this context, neladenoson bialanate holds promise as a potentially hemodynamically neutral therapy for HF that could simultaneously improve cardiomyocyte energetics, calcium homeostasis, cardiac structure and function, and long-term clinical outcomes when added to background therapies.




## 3.2 Partial adenosine A1 receptor agonism in heart failure

The failing heart is characterized by abnormal mitochondrial structure and function including hyperplasia and reduced organelle size, poor organelle respiration, reduced mitochondrial membrane potential, opening of membrane permeability pores, and reduced rates of adenosine triphosphate (ATP) synthesis and thereby reduced energy supply in cardiomyocytes in HFrEF and HF with preserved ejection fraction (HFpEF) (14-20). Additionally Ca<sup>2+</sup> handling is disturbed and SERCA<sub>2a</sub> protein levels are decreased in HF (21). This changes the contraction / relaxation coupling in cardiomyocytes and leads to an intracellular calcium overload in the heart. Furthermore, systemic metabolic impairments in the skeletal muscle are increasingly recognized as contributing both to symptoms (muscle weakness, exercise limitation) and disease progression in HF (22). Preclinical studies have demonstrated that myocardial energy metabolism and utilization as well as calcium homeostasis are improved by the partial adenosine A1 receptor agonist capadenoson (15, 23). In the heart failure standard dog model, treatment with this drug showed fast improvement of cardiac energetics (ATP synthesis) via mitochondrial effects. Capadenoson further improved SERCA<sub>2a</sub> activity, leading to decreased intracellular calcium overload (15).

The prevalence of coronary artery disease (CAD) is high in patients with HFrEF and HFpEF and associated with greater deterioration in ventricular function and increased mortality (24, 25) based mainly on ischemia driven injury of cardiac tissue. The primary physiological undertaking of adenosine is to preclude tissue injury and promote repair in response to stress mainly through adenosine A1 receptor (A1R) activation. Preclinical data showed cardioprotection from ischemia-induced injury by preconditioning and improvement of endothelial function in animal models with partial A1R agonists including capadenoson (15, 26, 27). Potential benefit of this targeted approach to the treatment of HF lies in the ability of partial A1R agonism to afford protection to the failing myocardium by limiting triggers of cell injury and death. Furthermore, the prevention of deterioration of myocardial ATP levels matching the ATP production to oxygen supply seems to be an important factor for cardioprotection. Especially patients with high risk for cardiac events (e.g. HF patients with diabetes, chronic kidney disease [CKD], advanced CAD) might benefit from A1R activation. Furthermore, excessive activation of the adrenergic nerve system is detrimental in HF

Furthermore, excessive activation of the adrenergic nerve system is detrimental in HF patients, inducing systemic vasoconstriction, increased sodium / water retention, and ventricular remodeling, all of which contribute to disease progression. Adenosine carries antiadrenergic properties that can protect the heart from adverse mechanical and metabolic stimulation from excessive catecholamine stimulation, thereby limiting ischemia. Activation of the A1R may also inhibit norepinephrine release from cardiac presynaptic nerves (28, 29). Conceivably, these effects may be important for preventing disease progression and further adverse remodeling, particularly in those with ischemic cardiomyopathy. Partial adenosine A1R agonism might offer a unique opportunity to selectively modulate the sympathetic control of cardiac function via presynaptic A1R activation and cAMP inhibition (28).

Heart failure is often associated with comorbidities like CKD and diabetes in HFrEF and HFpEF patients (30). Renal effects of adenosine A1R activation lead to vasoconstriction of the afferent arterioles in the kidneys (31) and thereby sodium retention and anti-diuretic effects. The effects were regarded as potential for renal benefit with adenosine antagonism in HF and led to large scale drug development programs with adenosine A1R antagonists, such




as rolofylline in patients with acute decompensated heart failure (ADHF). But the Phase III trial failed to show any renal protection. Instead, higher rates of persistent renal impairment, seizure and stroke were noted in the rolofylline group (32, 33). In contrast, an A1R agonist shows reno-protective effects in preclinical models of ischemia-induced renal injury (34). Increased plasma levels of free fatty acids (FFAs) are often found in patients with HF (35, 36) and result in an increase of insulin resistance and might be involved in the deterioration of heart function. A1R agonists can reduce plasma levels of FFAs in humans as shown in clinical trials (37). Furthermore, FFAs act as substrate for the energetic metabolism in the heart. HF is characterized by an added reliance on fatty acid oxidation, with downregulation of myocardial glucose transporters (38, 39). These changes characterize the transition of the failing heart to a fetal metabolic phenotype and gene profile, an adaptation that can further promote HF progression (38-40). Animal studies suggest that partial A1R agonist capadenoson can augment expression of the GLUT-1 and GLUT-4 glucose transporters to near normal levels (15). Moreover, therapy with capadenoson has also been associated with normalization of protein levels that mediate fatty acid oxidation (15). Thus, A1R agonism appears capable of partially correcting derangements in cardiac substrate utilization and restoring a physiologic metabolic profile in HF.

Previous attempts to address the A1 receptor, while offering potential therapeutic benefits, were limited by undesirable side effects that include bradycardia, atrioventricular blocks, sedation and antidiuretic effects. Furthermore, adenosine-like A1R agonists often have the drawback of a short half-life and low bioavailability making them not suitable for chronic oral therapy.

In contrast, partial adenosine A1 agonists may be used to modulate and trigger primarily favorable pharmacological responses for HF therapy, such as cardio- and renoprotection. A partial agonist is a low efficacy ligand, which elicits only a submaximal response from the receptor in contrast to a full agonist, even when all receptors are occupied. A partial agonist is expected to result in a robust signal response only in tissues with relative high receptor reserve, whereas a full agonist will elicit a robust signal also in tissue with a low receptor reserve. Thus, partial agonists are useful for achieving high selectivity for the target organ / tissue and minimizing toxicity and effects in non-target tissues (e.g. neurological effects, undesired kidney effects, AV conduction abnormalities). Hemodynamic effects evoked by A1R activation seem to have a lower receptor reserve in e.g. the AV node compared to cardioprotective effects. Furthermore, partial adenosine A1R agonists might induce less receptor desensitization than full agonists and be ideal for chronic treatment (41).

#### 3.3 Neladenoson bialanate

Neladenoson bialanate (BAY 1067197, which is the free base of the hydrochloride BAY 86-8901) is the pro-drug of the pharmacologically active compound BAY 84-3174, a highly potent and selective non-adenosine like partial adenosine A1 receptor agonist suitable for once daily oral use.

Pharmacological actions seem to be at least partly based on an acute restoration and improved utilization of myocyte energetics (ATP production within the mitochondria), and chronic improvement of calcium handling by restoration of SERCA<sub>2a</sub> protein levels, which result in protection of cardiac function and improvement of contraction / relaxation coupling. These effects were seen after a short treatment period of one week in nonclinical models. In




addition, neladenoson bialanate was characterized regarding mitochondrial function in isolated cardiomyocytes from normal and HF dogs (EF ~30%) produced by intracoronary microembolization as described in Sabbah et al (42). Neladenoson bialanate improved mitochondrial function (respiration, ATP synthesis, ATP / adenosine diphosphate [ADP] ratio, cytochrome c-dependent cyclooxygenase activity, membrane potential, and mitochondrial permeability transition pore opening) significantly and dose dependently in HF cardiomyocytes but had no effect on normal cardiomyocytes.

Nonclinical data showed that neladenoson bialanate is cardio- and renoprotective at doses lower than needed to elicit the clinically relevant undesirable effects on heart rate, AV-conduction, blood pressure, renal function and the central nervous system.

In animal models and clinical studies in healthy volunteers, neladenoson bialanate significantly reduces plasma levels of free fatty acids vs. placebo. Abnormal energetic activity in heart failure correlates inversely with plasma free-fatty-acid concentrations. The excess of fatty acids may adversely affect the myocardium and in HF may be associated with uncoupled respiration (43).

Further details can be found in the investigator's brochure (IB), which contains comprehensive information on the study drug. The IB in its most current version is available in the study file.

# 3.4 Rationale of the study

The main limitations of using full A1R agonists in cardiovascular indications such as HF are undesired cardiac effects, such as bradycardia and higher degree AV block as well as negative cardiac inotropy and dromotropy. In contrast, preclinical data show that the partial adenosine A1R agonist neladenoson bialanate can be used to modulate and trigger primarily favorable pharmacological responses for HF therapy and avoid undesired effects such as AV conduction abnormalities and higher degree AV Block. Nevertheless, based on the mode of action, there are theoretical concerns particularly with regard to undesired effects, such as bradycardia and higher degree AV block for an A1R agonist, which might be aggravated by concomitant use of standard heart failure therapy.

The purpose of this clinical trial is to assess the safety, tolerability and the pharmacokinetic and pharmacodynamic response of 20 weeks' treatment with neladenoson bialanate compared to placebo in patients with chronic HFrEF on standard therapy for HF and to find the optimal dose for a further Phase III trial.

# 4. Study objectives

The objective of the study is to find the optimal dose of neladenoson bialanate for the Phase III trial by detecting and characterizing a significant dose-response relationship in the two primary efficacy endpoints, absolute change from baseline in LVEF and log-transformed NT-proBNP at 20 weeks, in patients with chronic heart failure with reduced ejection fraction (HFrEF), and by characterizing the safety, tolerability and pharmacodynamic effects of the compound when given in addition to standard therapy for HFrEF.

An exploratory objective is to further assess pharmacokinetic parameters and blood and urine biomarkers.

For variables please see Section 10.3.1.




# 5. Study design

# 5.1 Design overview

Study 15128 is a randomized, double-blind, placebo-controlled, parallel group, multicenter, Phase II study. Figure 5–1 displays the overall study design.

Run-in Follow up Treatment placebo Eligibility check, baseline assessments, randomization events / hospitalizations 5 mg CF, eligibility check 10 mg End of treatment Safety follow-up 20 mg 30 mg 40 mg 2 W 2 W 4 W 8 W 12 W 20 W 26 W 19 W 24 W 0 W -1 Visit 3. Visit 4 Visit 5 Visit 6 Phone call Visit 7 Visit 9 Visit 8 Visit 1 Visit 2 phone call phone call

Figure 5-1: Study design overview

Abbreviations: CV = cardiovascular; ICF = informed consent form; W = week

Approximately 384 patients from approximately 90 study centers worldwide will be randomized to one of the active treatment dose arms or placebo, in addition to standard of care heart failure therapy (for details see Section 7).

The study will comprise a 1-week run-in period, 20-week treatment period, and a 6-week follow-up period (27 weeks total).

Patients will have site visits at weeks -1, 0 (baseline), 4, 8, 12, 20 (end-of-treatment visit) and 24 (safety follow-up visit). In addition, 2 phone calls at weeks 2 and 26 will be made to assess patients' safety, and one additional phone call - to remind the patients of AVIVO self-application at Week 19.

LVEF will be measured by echocardiography at baseline and end of treatment, NT-proBNP will be measured at baseline, Week 4 and end of treatment. Safety will be monitored throughout the study. PK samples will be taken from all patients at dedicated time points. Additional biomarkers reflecting the pharmacodynamic activity of the drug will be examined, as well as candidate biomarkers that may predict drug response.

For detailed visit descriptions and rules for patients who discontinue study treatment earlier, please see Sections 9.1 and 9.2.

The anticipated duration of the study as a whole is approximately 19 months: this includes an anticipated recruitment period of 13 months followed by a run-in period of 1 week, a treatment period of 20 weeks and a follow-up period of 6 weeks after enrollment of the last patient into the trial.




## 5.2 Primary variables

- Absolute change from baseline in left ventricular ejection fraction (LVEF; %) after 20 weeks measured by echocardiography.
- Absolute change from baseline in log-transformed NT-proBNP (pg/mL) after 20 weeks, i.e., log-transformed NT-proBNP at Week 20 minus log-transformed NT-proBNP at baseline.

For secondary and other variables please see Section 10.3.1.

# 5.3 Justification of the design

This section was changed in Amendment 2, see Section 15.1 for details.

A parallel group design was chosen to compare five different once-daily dose regimens and one placebo arm to find the best dose for Phase III. Placebo control is used to control for observer and subject bias, and randomization - to control for assignment bias. Based on Phase I data in healthy volunteers and Phase II data in heart failure patients, a sequential dose escalation design was not deemed necessary for neladenoson bialanate since the safety profile of the compound could be verified in dose ranges up to 40 mg. Evidence of A1R target engagement could already be achieved in different tissues across different clinical trials with 20 mg neladenoson bialanate. The dose range around 20 mg (5, 10, 30 and 40 mg) is to ensure different data points to feed the MCP-Mod predefined models and potential unforeseen variances. The doses studied will ensure a strong dose recommendation moving forward into phase III. Safety of the subjects in this parallel study design will be closely monitored by a Data Monitoring Committee (DMC).

# 5.4 End of study

The end of the study as a whole will be reached as soon as the last visit of the last patient has occurred in all centers in all participating countries (EU and non-EU).

# 6. Study population

#### 6.1 Inclusion criteria

Patients must meet all of the following inclusion criteria to be included in the study:

- 1. Men or women aged 18 years and older
- 2. Diagnosis of chronic heart failure (CHF), NYHA class II-IV, LVEF  $\leq$  35% assessed by any imaging modality (e.g. echocardiography, cardiac magnetic resonance, cine levocardiography) within 6 months prior to run-in: if several values are available the last assessment of LVEF should be  $\leq$  35%.
- 3. One of the following (or both),
  - a) Worsening CHF requiring hospitalization or an unscheduled outpatient visit in the last 3 months, both requiring initiation or intensification of heart failure therapy and with either:
    - o BNP  $\geq$  100 pg/mL or NT-proBNP  $\geq$ 400 pg/mL (sinus rhythm) or




 $\circ$  BNP  $\geq$  300 pg/mL or NT-proBNP  $\geq$ 1200 pg/mL (atrial fibrillation) AND/OR

- b) at any time in the past 4 weeks one of:
  - o BNP  $\geq$  300 pg/mL or NT-proBNP  $\geq$  1200 pg/mL (sinus rhythm)
  - o BNP  $\geq$  600 pg/mL or NT-proBNP  $\geq$  2400 pg/mL (atrial fibrillation)

For patients on treatment with angiotensin receptor-neprilysin inhibitors (ARNIs), e.g. Entresto only NT-proBNP values can be used to assess eligibility.

4. Written informed consent signed before any study-specific procedure

## 6.2 Exclusion criteria

This section was changed in Amendment 2, see Section 15.1 for details.

Patients who meet any of the following exclusion criteria will be excluded from the study:

- 1. Acute de-novo heart failure
- 2. Requirement of any of the following 48 hours prior to randomization:
  - o IV vasodilating drugs (e.g. nitrates, nitroprusside)
  - o IV natriuretic peptides (e.g. nesiritide, carperitide)
  - o IV positive inotropic agents
  - IV diuretics
  - o IV antibiotics
  - Mechanical support (e.g. intra-aortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device)
- 3. Any cause of chronic heart failure other than ischemic cardiomyopathy and idiopathic dilated cardiomyopathy
- 4. Known clinically significant persistent coronary ischemia based on medical history, preexisting or current exercise testing
- 5. Occurrence of any of the following within 3 months prior to randomization:
  - Myocardial infarction
  - o Hospitalization for unstable angina
  - o Stroke or transient ischemic attack
  - Coronary artery bypass graft (CABG)
  - o Percutaneous coronary intervention (PCI)
  - o Implantation of a cardiac resynchronization therapy device (CRTD)
  - Carotid angioplasty




- 6. PCI, CABG or implantation of a CRTD planned between randomization and end of study
- 7. Sustained ¹ systolic blood pressure ≤ 90 mmHg and / or signs and symptoms of hypotension prior to randomization
- 8. Sustained ¹ systolic blood pressure ≥ 160 mmHg
- 9. Sustained <sup>1</sup> bradycardia with heart rate < 50 beats/minute or tachycardia with heart rate > 100 beats/minute prior to randomization
- 10. Known clinically relevant ventricular arrhythmias (sustained ventricular tachycardia, ventricular flutter or fibrillation) within 3 months prior to consent based on either medical history or ICD-testing results (if applicable)
- 11. Clinically relevant permanent or intermittent AV-block ≥ grade II in patients without a permanent pacemaker or ICD / CRTD
- 12. Severe valvular disease with indicated or planned valve repair / replacement
- 13. Listing for heart transplantation and / or anticipated implantation of a ventricular assist device
- 14. Severe pulmonary disease with any of the following:
  - o Requirement of continuous (home) oxygen or
  - o History of chronic obstructive pulmonary disease ≥ GOLD III or
  - Use of systemic corticosteroids
- 15. Asthma bronchiale with any of the following:
  - o Symptoms not well-controlled within the past 6 months or
  - o Ever intubated or in an intensive care unit for asthma
- 16. Anemia with hemoglobin < 10 g/dL within 3 months prior to randomization. If several values are available the latest result should be used.
- 17. Body mass index (BMI) > 40 kg/m<sup>2</sup> at randomization or a history of poor quality LVEF measurement by echocardiography
- 18. Estimated glomerular filtration rate (eGFR) < 30 mL/min/1.73 m<sup>2</sup> calculated by Modification of Diet in Renal Disease (MDRD) formula within 3 months prior to randomization (see Appendix 16.1). If several values are available the latest result should be used.
- 19. Hepatic insufficiency classified as Child-Pugh B or C (see Appendix 16.2), or any of the following:
  - Primary biliary cirrhosis (PBC)
  - o Primary sclerosing cholangitis
  - o PBC-autoimmune hepatitis overlap syndrome

\_

<sup>&</sup>lt;sup>1</sup> At two consecutive visits




- 20. Concomitant use of any of the following therapy that cannot be discontinued:
  - Moderate or strong CYP3A4 inhibitors (Of note: grapefruit is a strong CYP3A4 inhibitor.)
  - CYP3A4 inducers
  - o Strong CYP2C8 inhibitors (Of note: clopidogrel is a CYP2C8 inhibitor)
  - o Theophylline
  - o Drugs having significant pre-systemic clearance via UGT1A1 in the intestine

Respective substances must be stopped at least 7 days before randomization.

- 21. Women of childbearing potential (women are considered of childbearing potential if they are not surgically sterile or postmenopausal, defined as amenorrhea for > 12 months)
- 22. Known current heavy alcohol consumption or the use of illicit drugs that, in the opinion of the investigator, may interfere with the patient's safety and / or compliance
- 23. Previous (within 30 days or 5 half-lives of the investigational drug, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s)
- 24. Previous assignment to treatment during this study
- 25. Any condition or therapy, which would make the patient unsuitable for the study, or life expectancy less than 12 months (e.g. active malignancy)
- 26. Close affiliation with the investigational site; e.g. a close relative of the investigator, dependent person (e.g. employee or student of the investigational site)
- 27. Known allergies, intolerance or hypersensitivities to the study treatment (active substance or excipients), adhesives or hydrogel

## 6.3 Justification of selection criteria

The selection criteria were chosen to exclude patients from the study who may potentially be exposed to specific risks after administration of the study drug, as well as patients with conditions that may have an impact on the aim of the study.

## 6.4 Withdrawal of patients from study

#### 6.4.1 Withdrawal

This section was changed in Amendment 2, see Section 15.1 for details.

An excessive rate of withdrawals (either patients discontinuing study medication or study withdrawal) can render the study non-interpretable. Therefore, un-necessary withdrawal of patients should be avoided and all efforts should be taken to motivate patients to comply with all the study specific procedures and to be followed until the end of the trial to detect the occurrence of cardiovascular events / assess vital status.

Before permanently discontinuing study medication (either initiated by the patient or the investigator) an interruption should be considered. Patients, who have temporarily discontinued study medication for any reason, should restart as soon as medically justified in the opinion of the investigator; the patient can re-start at any time before the end of treatment




(EOT) visit. In addition, patients should not be withdrawn from the study drug or from the study solely due to reaching a potential cardiovascular event.

All patients who permanently discontinue study medication should come in for the EOT / premature discontinuation visit as soon as possible after discontinuation of the study medication and the safety follow-up visit 4 weeks after the last dose. In addition, they will be contacted by the investigator via the scheduled Week 26 phone call to assess occurrence of cardiovascular events.

The investigator should show due diligence and explore all possible options to reach a patient who fails to return to a visit. The site must document all attempts to try to contact the patient in the medical records / source documents.

In order to avoid loss-to-follow-up, the investigator should ask the patient at the study start for the contact details of a relative or friend who can be contacted in case the patient cannot be reached.

Patients should not be withdrawn from follow-up unless the patient explicitly withdraws consent to be contacted. All efforts should therefore be made to minimize the number of patients who withdraw such consent as, in general, no further information on cardiovascular events and survival status may be collected after that point.

#### Withdrawal criteria

Patients *must* be withdrawn from the study if any of the following occurs:

• At their own request or at the request of their legally acceptable representative. At any time during the study and without giving reasons, a patient may decline to participate further. The patient will not suffer any disadvantage as a result.

Patients *may* be withdrawn from the study if any of the following occurs:

- If, in the investigator's opinion, continuation of the study would be harmful to the patient's well-being.
- At the specific request of the sponsor and in liaison with the investigator (e.g. obvious non-compliance, safety concerns).
- If any investigational drug other than the study drug is used during the study period.

Depending on the time point of withdrawal, a withdrawn patient is referred to as either "screening failure" or "dropout" as specified below.

### Screening failure

A patient who, for any reason (e.g. failure to satisfy the selection criteria), terminates the study before randomization is regarded a "screening failure".

Re-screening is allowed once and only in the following cases:

- The patient had successfully passed the screening procedures, but could not start subsequent treatment on schedule.
- Initial screening occurred too early to complete the required washout period for prohibited substances.




In any case, the investigator has to ensure that the repeated screening procedures do not expose the patient to an unjustifiable health risk. For re-screening, the patient must sign a new informed consent form, even if its version was not changed after the patient's previous screening. In the event of re-screening the patient will be assigned a new patient identification number.

#### **Dropout**

A patient who discontinues study participation prematurely for any reason is defined as a "dropout" if the patient has already been randomized whether or not any study medication was taken.

## **General procedures**

In all cases, the reason for withdrawal must be recorded in the CRF and in the patient's medical records.

The patient may object to the generation and processing of post-withdrawal data as specified in Section 13.4.

Details for the premature termination of the study as a whole (or components thereof) are provided in Section 12.

### 6.4.2 Replacement

Randomized patients who drop out or withdraw prematurely will not be replaced.

#### 6.5 Patient identification

The patient number is a 9-digit number consisting of:

Digits 1 to 5 = Unique center number

Digits 6 to 9 = Current patient number within the center

#### 7. Treatments

### 7.1 Treatments to be administered

Patients will receive either active treatment with neladenoson bialanate or placebo; treatment assignment is described in Section 7.3. Patients will be instructed to take two study tablets once daily, preferably in the morning, over a period of 20 weeks. On visit days, the study drug should be taken as specified in Table 9–1. The study drug should be taken with a glass of water, and can be taken with or without food. There will be no dose modifications; patients will stay on the dose which they were randomized to. For guidance regarding drug discontinuation please see Section 6.4.1.

This treatment will be in addition to patients' regular heart failure treatments (see Section 8.1.2).

## 7.2 Identity of study treatment

Three different "BAY-numbers" are used within this document, corresponding to three different chemical appearances of neladenoson bialanate:




**BAY 1067197** is a pro-drug. BAY 1067197 represents the "pharmaceutical principle" of neladenoson bialanate, and thus this BAY number is used when generally speaking about neladenoson bialanate. Present dosages refer to BAY 1067197.

**BAY 86-8901** is the hydrochloride salt of BAY 1067197. BAY 86-8901 is used to formulate the immediate release tablets to be administered to study patients. This BAY number is used when speaking about the oral preparation of neladenoson bialanate.

BAY 1067197 cannot be found in measurable concentrations, or only at very low concentrations in the blood plasma. Orally administered drug is converted by ester cleavage into the active metabolite **BAY 84-3174**, which is responsible for the pharmacodynamic effects. BAY 84-3174 is used in the context of plasma pharmacokinetic data measurements.

Details of BAY 1067197 are given in Table 7–1; details of placebo are given in Table 7–2. For more information please refer to the latest available version of the investigator's brochure.

Table 7-1: Identity of neladenoson bialanate (BAY 1067197)

| Sponsor's internal reference number | BAY 1067197 |
|---|---|
| Formulation | Pink coated tablets |
| Galenical form | Round biconvex, diameter 8 mm Markings: One side PT; Other side blank |
| Composition | Active ingredient: neladenoson bialanate, 2-{4-[2-({[2-(4-chlorophenyl)-1,3-thiazol-4-yl]methyl}sulfanyl)-3,5-dicyano-6-(pyrrolidin-1-yl)pyridin-4-yl]phenoxy}ethyl L-alanyl-L-alaninate |
| | Empirical formula: C <sub>35</sub> H <sub>34</sub> Cl N <sub>7</sub> O <sub>4</sub> S <sub>2</sub> * HCl |
| | Molecular mass: 716.29 + 36.46 [g/mole] |
| | Excipients: Lactose anhydrous, Crospovidone and magnesium stearate |
| | Coating: Lacquer pink (Opadry Pink 02A34744) |
| Strength | 5 mg,10 mg and 20 mg |
| Packaging | Blister |

### Table 7-2: Identity of placebo

| Formulation | Pink coated tablets |
|---|---|
| Galenical form | Round, biconvex, diameter 8 mm |
| | Markings: One side PT; Other side blank |
| Composition | lactose monohydrate, cellulose microcrystalline and magnesium stearate |
| | Coating: Lacquer pink (Opadry Pink 02A34744) |
| Packaging | Blister |

#### **Storage requirements**

Study drug will be stored at the investigational sites according to the label requirements in a place inaccessible to unauthorized personnel, i.e. in a locked cabinet.

All study drugs will be labeled according to the requirements of local law and legislation. Label text will be approved according to the sponsor's agreed procedures, and a copy of the labels will be made available to the study site upon request.




For all study drugs, a system of numbering in accordance with all requirements of GMP will be used, ensuring that each dose of study drug can be traced back to the respective bulk batch of the ingredients. Lists linking all numbering levels will be maintained by the sponsor's clinical supplies quality assurance group.

A complete record of batch numbers and expiry dates of all study treatment as well as the labels will be maintained in the sponsor's study file.

# 7.3 Treatment assignment

The intention is to randomize approximately 384 subjects to the doses 5 mg, 10 mg, 20 mg, 30 mg, 40 mg of neladenoson bialanate, and placebo according to an allocation ratio of 1:2:2:2:2:3, respectively.

At the baseline visit, the investigator will first perform all required pre-treatment examinations and will then randomize the qualified patients to one of the six treatment arms.

The randomization will be stratified by atrial fibrillation (AF): yes vs. no.

Enrollment into the AF stratum may be stopped (after the discussion between the sponsor and the Steering Committee) when the AF stratum constitutes 30% of the total expected enrollment.

The randomization lists will be provided by Bayer's Global Randomization Management Group. Randomization will be done using an interactive voice / web response system (IxRS).

A handbook describing how to use the IxRS will be provided to each study site.

## 7.4 Dosage and administration

For dosage and administration please refer to Section 7.1.

## 7.5 Blinding

This section was changed in Amendment 2, see Section 15.1 for details.

All patients will receive the same number of tablets (only active, combination of active and placebo or only placebo, depending on the treatment arm) to maintain the blind (Table 7–3).

Table 7-3: Assignment of tablets to dose groups

| Treatment arm/<br>Formulation | 5 mg | 10 mg | 20 mg | 30 mg | 40 mg | Placebo |
|---|---|---|---|---|---|---|
| 5 mg | 1 | 0 | 0 | 0 | 0 | 0 |
| 10 mg | 0 | 1 | 0 | 1 | 0 | 0 |
| 20 mg | 0 | 0 | 1 | 1 | 2 | 0 |
| Placebo | 1 | 1 | 1 | 0 | 0 | 2 |
| Total tablets/day | 2 | 2 | 2 | 2 | 2 | 2 |

The following parties will be unblinded: sponsor's IxRS and Medication Manager, Clinical Supply Manager and Clinical Pharmacometrics analyst (who will be provided with a randomization list for selected bioanalyses of the active metabolite BAY 84-3174 in plasma), the drug supply's Project Manager, and the DMC.




For all other sponsor's study personnel, the Steering Committee and the Clinical Events Committee (CEC) the blinding will be strictly kept.

In compliance with applicable regulations, in the event of a SUSAR (see Section 9.6.1.5) related to the blinded treatment, the patient's treatment code will usually be unblinded before reporting to the health authorities, ethic committees and investigators (see Section 9.6.1.4). For exceptions please see Section 9.6.1.4.

#### **Emergency unblinding by the investigator**

In the event of emergency, and where knowledge of assigned treatment allocation is required for the acute treatment strategy, the investigator may unblind the case. Unblinding will be handled in IxRS.

The occurrence of SAEs should not routinely precipitate the immediate unblinding. The investigator is required to promptly document and explain to the sponsor any premature unblinding (e.g. unblinding due to an SAE) of the study drug. The investigator should report unblinding of treatment to the EC / IRB according to the EC / IRB's requirements.

# 7.6 Drug logistics and accountability

All study drugs will be stored at the investigational site in accordance with GCP and GMP requirements and the instructions given by the clinical supplies department of the sponsor (or its affiliate), and will be inaccessible to unauthorized personnel. Special storage conditions and a complete record of batch numbers and expiry dates can be found in the sponsor's study file; the site-relevant elements of this information will be available in the investigator site file. On the day of receipt, the responsible site personnel will confirm receipt of study drug via IxRS. The personnel will use the study drug only within the framework of this clinical study and in accordance with this protocol. Receipt, distribution, return and destruction (if any) of the study drug must be properly documented according to the sponsor's agreed and specified procedures.

Written instructions on medication destruction will be made available to affected parties as applicable.

#### 7.7 Treatment compliance

To monitor compliance, the investigator will be required to document drug dispensing for each patient. Overall compliance with study drug intake should be between 80% and 120% of the scheduled dose at the end of study drug treatment. The date of dispensing the study drug to the patient will be documented.

Study drug will be dispensed according to the schedule provided in Section 9.1.

Patients will return at scheduled visits or at the premature discontinuation / EOT visit, if applicable, with all remaining unused study drug, when accountability will be determined for all tablets. To facilitate this, patients must be instructed to return all of the study drug packaging including unused study drug and empty packaging.

Any discrepancies between actual and expected amount of returned study medication must be discussed with the patient at the time of the visit, and any explanation must be documented in the source records.




# 8. Non-study therapy

# 8.1 Prior and concomitant therapy

### **8.1.1** Prohibited concomitant medication

This section was changed in Amendment 2, see Section 15.1 for details.

Concomitant therapy with any of the following drug classes is prohibited:

- Moderate or strong CYP3A4 inhibitors (Of note: grapefruit is a also strong CYP3A4 inhibitor)
- CYP3A4 inducers
- Strong CYP2C8 inhibitors (Of note: clopidogrel is a strong CYP2C8 inhibitor)
- Theophylline
- Drugs having significant pre-systemic clearance via UGT1A1 in the intestine

Respective substances must be stopped at least 7 days before randomization and can only be started 6 weeks after the last intake of study drug. A list of prohibited medications will be provided to the investigators.

If a prohibited concomitant medication (e.g. moderate / strong CYP3A4 inhibitor) is used during the study conduct, the study drug should be interrupted immediately and restarted as soon as possible, when the prohibited medication has been stopped. Prior to re-starting the study drug, a washout period of at least two days after discontinuation of the prohibited medication should be adhered to.

# 8.1.2 Permitted therapy

This section was changed in Amendment 2, see Section 15.1 for details.

- In accordance with standard local or international heart failure guidelines, all patients should be on standard HF therapy (an ACEi or ARB, beta-blockers, MRA, ARNI, as applicable), unless contraindicated or (to the investigator's knowledge) not tolerated
- Concomitant therapy of comorbidities is allowed unless listed in the prohibited medication section.

During the treatment period the background medications should be kept stable and changes in treatment should be based on clinical need.

Neladenoson bialanate is a weak Breast Cancer Resistance Protein (BCRP) inhibitor. The risk of clinically relevant drug—drug interactions at doses up to 40 mg BAY 1067197 due to inhibition of BCRP is regarded as low, but cannot be excluded (BCRP substrates are atorvastatin, simvastatin, rosuvastatin, fluvastatin, methotrexate, etc.; a list of BCRP substrates will be made available to the investigators).

If neladenoson bialanate is given concomitantly with other drugs that may increase the exposure of BCRP substrates, the respective drug labels should be consulted.

All concomitant medication will be documented in the eCRF.




# 8.2 Post-study therapy

The investigator must provide follow-up medical care for all patients who complete the study or who are prematurely withdrawn from the study, or must refer them for appropriate ongoing care, as required.

Study medication will not be available to patients after completion of the study.

# 9. Procedures and variables

# 9.1 Tabular schedule of evaluations

This section was changed in Amendment 2, see Section 15.1 for details.




Table 9–1: Schedule of evaluations

| Study period | Run<br>-in | | varaat | | ment <sup>a</sup> | | | EOT /<br>PDV | Safety<br>FU | | o p |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit number | 1 | 2 | 3 | 4 | 5 | 6 | | 7 | 8 | 9 | nle |
| Visit type | site | site | 2 | site | site | site | <b>a</b> b | site | site | * | Unscheduled |
| Week | -1 | W0 | W2 | W4 | W8 | W12 | W19 | W20 <sup>a</sup> | <b>W24</b> <sup>c</sup> | W26 <sup>a</sup> | sch |
| Day and allowed deviations | | 0+2 | 14±2 | 28±2 | 56±2 | 84±2 | 133-2 | 140±2 | 168 ±2 | 182+7 | 'n |
| Day and anomed deviations | <u> </u> | Pre-rand. | | | LOGIE | 0.112 | 1.00 = | 17012 | 100 12 | 102.7 | |
| Signed informed consent | • | i io iana. | | | | | | | | | |
| Inclusion / exclusion | • | • | | | | | | | | | |
| KCCQ | | • | | • | | • | | • | | | |
| EQ-5D-5L | | • | | | | | | • | | | |
| | _ | • | | | | | | • | | | |
| Demographic data | • | | | | | | | | | | |
| Medical and surgical history | | • | | | | | | | | | |
| Smoking & alcohol history | | • | | | | | | | | | |
| Caffeine & chocolate consumption | | • | | | | | | • | | | |
| Physical exam | | • | | • | • | • | | • | ● <sup>d</sup> | | • |
| Height | | • | | | | | | | | | |
| Weight | | • | | • | • | • | | • | • | | • |
| 12-lead ECG | | • | | | | • | | • | | | |
| NYHA class | | • | | • | • | • | | • | • | | • |
| Blood pressure and heart | _ | _ | | _ | _ | _ | | _ | _ | | |
| rate | • | • | | • | • | • | | • | • | | <u> </u> |
| Adverse events | • | • | • <sup>e</sup> | • | • | • | | • | • | ● <sup>e</sup> | • |
| Concomitant medication | • | • | • | • | • | • | | • | • | • | • |
| AVIVO application, worn for 7 days | • | • | | | • | f | • | | | | |
| Collection of AVIVO device | | • | | • | | • | | • | | | |
| Echocardiography (central) | | • | | | | | | • | | | |
| Randomization via IxRS | | • | | | | | | | | | |
| Transcomization via ixivo | | post-rand | l | | <u> </u> | | | | | | |
| Laboratory (central lab) | | poor raile | • | | | | | | | | |
| Blood sample for safety | | pre-<br>dose | | | | • | | • | • | | • |
| PK sample (exact time to | | 2h post- | | pre- | pre- | ~2h & 4h | | 1 day | | | |
| be documented) <sup>g</sup> | | dose | | dose | dose | post-dose | | post-dose | • | | |
| Blood sample for | | pre- | | | | | | • | ● <sup>h</sup> | | |
| biomarkers | | dose | | • | | | | • | • | | |
| Urine sample for | | pre-<br>dose | | • | | | | • | | | |
| biomarkers Study drug i | | 4030 | <u> </u> | ı | | | | | | | |
| Study drug intake at the | | | | | | | | | | | |
| site | | • | | • | • | | | | | | |
| Study drug intake before the visit | | | | | | ~2h<br>before | | 1 day<br>before | | | |
| Patients to remember time | | | | day | day | - | | day of last | | | |
| of the study drug intake | | | | | before | • | | dose | | | |
| Dispense contact card | • | | | | | | | | | | |
| Dispense study drug | | • | | • | • | • | | | | | |
| Collect unused study drug | | | | • | • | • | | • | | | |




#### Table 9-1: Schedule of evaluations (continued)

Abbreviations: ECG = electrocardiogram; EOT = end of treatment; EQ-5D-5L = EuroQol Group 5-dimensional, 5-level questionnaire; FU = follow-up; h = hour(s); IxRS = interactive web/voice response system; KCCQ = Kansas City Cardiomyopathy Questionnaire; NYHA = New York Heart Association; PDV = premature discontinuation visit; post-rand. = post-randomization; PK = pharmacokinetics; prerand. = pre-randomization; W = week

- a For patients who discontinue study medication prematurely:
  - EOT / premature discontinuation visit must be performed as soon as possible after discontinuation of the study drug.
  - Safety FU visit must be scheduled 4 weeks after the last dose (± 2 days).
  - Week 26 follow-up call will be made 26 weeks after the start of treatment (+7 days).
- b Phone call to remind patients to self-apply AVIVO device. The phone can be made up to 2 days before Week 19, but not later than Week 19, to have 7 days of data for evaluation at the Week 20 visit.
- c Safety FU visit is relative to the last dose of study medication and is 4 weeks after the last dose.
- d Targeted physical examination based on symptoms
- e If there is an AE reported during a phone call, the investigator, at his / her discretion, may ask the patient to come for an unscheduled visit at the patient's earliest convenience (Section 9.2.11).
- f At Visit 6 (Week 12) the site will hand over AVIVO device to patients for self-application at Week 19 and instruct them how to apply the device.
- g **At Visit 2**: One PK sample will be drawn not earlier than 2 hours and not later than 6 hours after the first dose of study medication. Exact time of the first dose must be recorded by the investigator.
  - **At Visits 4 and 5**: One PK sample at each of the visits will be drawn pre-dose. Patients must not take study medication before the visit but should remember exact time of the previous dose.
  - At Visit 6: Two PK samples will be drawn post-dose
    - 1. 2 hours after the study drug intake (range 1:30 hour to 3:29 hours)
    - 2. 4 hours after the study drug intake (range 3:30 hours to 5:30 hours)

The minimum time between the two samples should be at least 1 hour.

Patients will be instructed to take the study drug about 2 hours before the visit and to remember the exact time. If a patient does not take the study drug before the visit, he / she can take it at the start of the visit, in which case PK sampling will occur as described above.

**At Visit 7**: One PK sample will be drawn 1 day after the last dose. Patients should remember the exact time of their last dose.

#### h Only NT-proBNP

i It is important that the patients remember the time of the tablet intake as precisely as possible (i.e. exact hour and minute) on the following days:

- 1. On the day before Visits 4 and 5
- 2. On the day of Visit 6
- 3. On the day of their last dose.

This information will be recorded in the patient's file. A phone call to remind the patients is recommended. Investigator must record the time of the dose when the study drug is taken at the site.




## 9.2 Visit description

This section was changed in Amendment 2, see Section 15.1 for details.

# 9.2.1 Visit 1 (Week -1, run-in)

- Confirm signed informed consent is available (Section 13.4)
- Allocate unique patient identification number (Section 6.5)
- Eligibility assessment (Sections 6.1 and 6.2)
- Demographic data collection and recording (Section 9.3.1)
- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- AVIVO device application, worn for 7 days (Section 9.6.3.5)
- Contact card dispensing

# 9.2.2 Visit 2 (Week 0, baseline)

At Visit 2 eligibility must be re-assessed before the patient is randomized to a treatment arm. Please note: laboratory eligibility criteria are based upon local and historical records, not central laboratory findings. Even retrospectively, central laboratory results from the baseline visit will not render a patient ineligible for the study. If a patient is not eligible for randomization, or withdraws for other reasons before randomization, he/she will be considered a screening failure even though the visit is not named a screening visit (for details see Section 6.4.1).

The following procedures will be performed **before randomization**:

- Review in/exclusion criteria and confirm patient eligibility
- Quality of life questionnaires (KCCQ and EQ-5D-5L), to be completed by the patient (Section 9.4.4)
- Medical and surgical history collection and recording (Section 9.3.2)
- Tobacco smoking and alcohol history collection and recording
- Assessment of caffeine-containing beverage and chocolate consumption during the previous 4 weeks
- Physical examination (Section 9.6.3.2)
- Weight and height measurement (BMI will be calculated automatically)
- 12-lead ECG (Section 9.6.3.3)
- NYHA class assessment (Section 9.4.3.2)
- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- Collection of AVIVO device applied at Visit 1 (Week -1)
- Echocardiography (Section 9.4.1)




• AVIVO device application, worn for 7 days (Section 9.6.3.5)

After all above procedures are done, the patient can be randomized via IxRS (Section 7.3).

The following procedures should be performed after randomization and before study medication intake:

- Blood sampling for safety (Section 9.6.3.1)
- Blood and urine sampling for biomarkers (Section 9.4.2)
- Study drug dispensing (Section 7.7)

The following procedures should be performed during and after study medication intake:

- Start of study medication (Section 7.1). The first dose of study medication will be taken after all previous procedures are completed; the time of intake should be recorded. The patients will be instructed to remember the time of medication intake as precisely as possible on selected days.
- PK sampling not earlier than 2 hours and not later than 6 hours after the first dose of study medication; exact time of PK sampling and drug intake is to be documented in the patient's file (Section 9.5)

# 9.2.3 Visit 3 (Week 2, phone call)

After 2 weeks of treatment ( $\pm$  2 days) the site personnel will call the patients to inquire about adverse events and to collect information on concomitant medications. If there is an AE reported during the phone call, the investigator may ask the patient to come for an unscheduled visit (Section 9.2.11). Information collected during the phone call must be recorded in the patient's medical records / source documents.

# 9.2.4 Visit 4 (Week 4)

- Quality of life questionnaire (KCCQ), to be completed by the patient (Section 9.4.4.1)
- Physical examination (Section 9.6.3.2)
- Weight measurement
- NYHA class assessment (Section 9.4.3.2)
- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- Collection of AVIVO device applied at Visit 2 (Week 0)
- Blood sampling for safety (Section 9.6.3.1)
- PK sampling (pre-dose). Please note: on this day the patients should not take the study medication before the visit but only after the PK sampling. Ideally, the study personnel should contact the subject prior to Visit 4 to remind them not to take the study drug as usual in the morning at home. The patient should remember the time of the previous study drug intake as precisely as possible. Exact time of PK sampling and drug intake is to be documented in the patient's file.



- Blood and urine sampling for biomarkers (Section 9.4.2)
- Study drug dispensing and unused study drug collection (Section 7.7)

# 9.2.5 Visit 5 (Week 8)

- Physical examination (Section 9.6.3.2)
- Weight measurement
- NYHA class assessment (Section 9.4.3.2)
- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- AVIVO device application, worn for 7 days (Section 9.6.3.5)
- Blood sampling for safety (Section 9.6.3.1).
- PK sampling (pre-dose). Please note: on this day the patients should not take the study medication before the visit but only after the PK sampling. Ideally, the study personnel should contact the subject prior to Visit 5 to remind them not to take the study drug as usual in the morning at home. The patient should remember the time of the previous study drug intake as precisely as possible. Exact time of PK sampling and drug intake is to be documented in the patient's file.
- Study drug dispensing and unused study drug collection (Section 7.7)

# 9.2.6 Visit 6 (Week 12)

- Quality of life questionnaire (KCCQ), to be completed by the patient (Section 9.4.4.1)
- PK sampling (Section 9.5):
  - Study drug is to be taken at home approximately 2 hours before the visit; it is important that the patients remember the time of study drug intake as precisely as possible; a phone call on the previous day to remind the patients is recommended. This information will be documented in the patient's file.
  - The first PK sample is to be taken approximately 2 hours after study drug intake (range 1:30 hour to 3:29 hours). Time of sampling should be precisely documented in the patient's file.
  - o The second PK sample is to be taken approximately 4 hours after study drug intake (range 3:30 hours to 5:30 hours). Time of sampling should be precisely documented in the patient's file.
  - o The minimum time between the two samples should be at least 1 hour.

If a patient does not take the study drug before the visit, he / she can take it at the start of the visit, in which case PK sampling will occur as described above.

- Physical examination (Section 9.6.3.2)
- Weight measurement
- 12-lead ECG (Section 9.6.3.3)




- NYHA class assessment (Section 9.4.3.2)
- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- Collection of AVIVO device applied at Visit 5 (Week 8)
- Handing-over AVIVO device to patients for self-application at Week 19 (Section 9.2.7) and instruction of patients how to apply the device
- Blood sampling for safety (Section 9.6.3.1)
- Study drug dispensing and unused study drug collection (Section 7.7)

# 9.2.7 Reminder phone call at Week 19

After 19 weeks of treatment (- 2 days) the site personnel will call the patients to remind them to self-apply the AVIVO device provided at Visit 6 (Week 12); if the device has not been provided at site, it should have been shipped to the patients. If there is an AE reported during the phone call, the investigator will have to make sure this is further assessed at the Week 20 visit or at an unscheduled visit prior to this.

Every effort should be made that the Week 20 visit at the site is conducted 7 days after the patient has applied the AVIVO device to have 7 days of data for evaluation. Accordingly, scheduling of Week 19 reminder-call and Week 20 visit should be aligned to achieve this. If the site prefers to have an on-site visit at Week 19 for the purposes mentioned above, an unscheduled visit (Section 9.2.11) can be conducted instead of the phone call (the patient's preference should also be considered). Information collected during the phone call must be recorded in the patient's medical records / source documents.

## 9.2.8 Visit 7 (Week 20, EOT or premature discontinuation)

The last dose of study drug should be taken the day before the visit. The patients should remember the time of the last dose as precisely as possible; this information will be recorded in the patient's file. It is recommended to make a reminder phone call to the patients on the previous day.

If a patient discontinues study treatment prematurely, this visit should be completed as soon as possible after the last dose.

- Quality of life questionnaires (KCCQ and EQ-5D-5L), to be completed by the patient (Section 9.4.4)
- Physical examination (Section 9.6.3.2)
- Weight measurement
- Assessment of caffeine-containing beverage and chocolate consumption during the previous 4 weeks
- 12-lead ECG (Section 9.6.3.3)
- NYHA class assessment (Section 9.4.3.2)




- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- Collection of AVIVO device applied at Week 19
- Echocardiography (Section 9.4.1)
- Blood sampling for safety (Section 9.6.3.1)
- PK sampling one day after the last dose (Section 9.5)
- Blood and urine sampling for biomarkers (Section 9.4.2)
- Unused study drug collection (Section 7.7)

# 9.2.9 Visit 8 (Week 24, safety follow-up)

If a patient discontinues study treatment prematurely this visit should be completed 4 weeks  $\pm 2$  days after the last dose.

- Physical examination (targeted examination based on symptoms) (Section 9.6.3.2)
- Weight measurement
- NYHA class assessment (Section 9.4.3.2)
- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- Blood sampling for safety (Section 9.6.3.1)
- PK sampling (Section 9.5)
- Blood sampling for NT-proBNP (Section 9.4.2)

## 9.2.10 Visit 9 (Week 26, phone call)

Twenty-six weeks after the start of study treatment the site personnel will call the patients to inquire about adverse events, including cardiovascular events, and to collect information on concomitant medications. For patients who discontinue study drug treatment early, the phone call will still be made 26 weeks after the start of study treatment. Information collected during the phone call must be recorded in the patient's medical records / source documents.

#### 9.2.11 Unscheduled Visit

If a patient experiences an adverse event for which the investigator determines a follow-up site visit is necessary (either before the next scheduled study visit or during the Week 26 phone call), then the following assessments will be performed:

- Physical examination (Section 9.6.3.2)
- Weight measurement
- NYHA class assessment (Section 9.4.3.2)




- Blood pressure and heart rate measurement (Section 9.6.3.4)
- Adverse events assessment (Section 9.6.1.3)
- Concomitant medication collection and recording (Section 8.1)
- Blood sampling for safety (Section 9.6.3.1)

# 9.3 Population characteristics

## 9.3.1 Demographic and vital signs

The following demographic and vital signs data will be collected and recorded in the eCRF:

- Year of birth
- Age (to be calculated by the investigator)
- Gender
- Race / ethnicity (collection may be restricted per local regulations)
- Weight
- Height

BMI will be calculated automatically.

### 9.3.2 Medical history

Medical history findings (i.e. previous diagnoses, diseases or surgeries) meeting all criteria listed below will be collected as available to the investigator:

- Start before signing of the informed consent
- Pertaining to the study indication
- Considered relevant to the study (e.g. cardiovascular and metabolic diseases)
- Considered relevant for the patient's study eligibility
- Related to concomitant medication

Detailed instructions on the differentiation between (i) medical history and (ii) adverse events can be found in Section 9.6.1.1.

## 9.3.3 Other baseline characteristics

In addition, the following baseline characteristics will be collected and recorded:

- Pre-defined medical history
- NYHA class
- Tobacco smoking history
- Alcohol consumption history
- Recent caffeine-containing beverage and chocolate consumption history




# 9.4 Efficacy

# 9.4.1 Echocardiography

Transthoracic echocardiography and tissue Doppler will be performed at the time points specified in Section 9.1. The readings will be assessed centrally. SBP, DBP, and HR will be measured during echocardiography in addition to acquisition of echo data. The following parameters (but not limited to) will be analyzed by the central reader:

- LV ejection fraction (LVEF, %)
- LV end-diastolic volume (LVEDV), LVEDV index (LVEDVI, calculated as LVEDV/BSA)
- LV end-systolic volume (LVESV), LVESV index (LVESVI, calculated as LVESV/BSA)
- LA size (LA diameter, area, volume index [LAVI, calculated as LAV/BSA])
- Lateral e' (early diastolic mitral annular relaxation velocity at the lateral mitral annulus by Tissue Doppler, TD)
- Septal e' (early diastolic mitral annular relaxation velocity at septal mitral annulus by TD), including calculation of average e'
- Global longitudinal strain (%)
- Pulmonary artery systolic pressure (PASP), estimated by tricuspid regurgitation velocity and inferior vena cava diameter, including its change with respiration, and hepatic vein flow in patients with tricuspid regurgitation
- Tricuspid annular plane systolic excursion (TAPSE), right ventricular (RV) s' (velocity of the tricuspid annular systolic excursion at the RV free wall by TD)
- Mitral regurgitation
- LV mass, LV mass index (calculated as LV mass/BSA)
- Wall thicknesses, incl. interventricular septum diameter (IVSD), posterior wall thickness (PWT), anteroseptal wall thickness (ASWT)
- E, A (if in sinus rhythm), calculation of E/A and E/e' (using lateral, septal, average e') ratios
- E-wave deceleration time (EWDT)
- Stroke volume (SV, calculated by LVEDV LVESV) and derived parameters, including SV index (SVI, calculated as SV/BSA), cardiac output (CO, calculated as SV\*HR), cardiac index (CI, calculated as CO/BSA), systemic arterial compliance (SAC, calculated as SV/PP), total peripheral resistance (TPR, calculated as MAP/CO\*80)
- Effective arterial elastance (Ea), estimated as end-systolic pressure (Pes) [Pes calculated as SBP times 0.9 (44)] divided by SV (SBP\*0.9/SV)

Final details of all echocardiography parameters to be measured and analyzed will be included in a separate echocardiography manual.




## 9.4.2 Biomarker investigations

This section was changed in Amendment 2, see Section 15.1 for details.

Biomarker investigations in the present study will include the biomarkers listed below.

# Mandatory (sampled at all time points):

- NT-proBNP (baseline disease status & efficacy)
- High sensitivity troponin T (hs-TNT) (baseline disease status)
- Cystatin C (baseline disease status & efficacy)
- Free fatty acid (FFA) (target engagement / mechanistic marker)
- Urine albumin-to-creatinine ratio (UACR)
- Hemoglobin A1c (HbA1c) (target engagement / mechanistic marker)
- Neutrophil gelatinase-associated lipocalin (NGAL) (baseline disease status & efficacy)

# Additional exploratory biomarker sampling:

- Soluble suppression of tumorigenicity-2 (sST2) (baseline disease status & efficacy)
- Galectin-3 (Gal-3) (baseline disease status & efficacy)
- Growth differentiation factor 15 (GDF-15) (baseline disease status & efficacy)
- Mid-regional pro-atrial natriuretic peptide (MR-proANP) (baseline disease status & efficacy)
- Copeptin (baseline disease status & efficacy)
- Osteopontin (OPN) (baseline disease status & efficacy)
- Tissue inhibitor of metalloproteinase-4 (TIMP-4) (baseline disease status & efficacy)
- Additional newly emerging HF or safety biomarkers

Blood sampling for biomarkers is scheduled for the time points as given in Section 9.1. All biomarkers will be measured using validated assay systems. Quality control (QC) and calibration samples will be analyzed concurrently with study samples. The results of the QC samples will be reported in a separate analytical report. Details on the collection, processing, storage and shipment of biomarker samples will be provided in separate documents (e.g. sample handling sheets or lab manual). Additional exploratory biomarkers sampling is to be used for research purposes to identify and / or verify biomarkers that are predictive or correlate with the efficacy / safety and the response in terms of tolerability of neladenoson bialanate. The analysis of exploratory biomarker may include the listed above exploratory biomarkers, safety biomarkers or new emerging HF biomarkers. Exploratory biomarker statistics may be reported separately. Exploratory biomarker analysis completed in the first year after the end of the study will be reported back to the investigator, if this provides additional meaningful information. Pure exploratory measures without an established interpretation might be withheld of reporting, considering that this will be of no value to the investigator or patient. The steering committee will provide guidance to the sponsor on reporting of exploratory biomarkers to investigators and patients.




In addition to the biomarkers listed above, other biomarkers deemed relevant to gain further knowledge about the pathomechanism of the disease or about the drug (i.e. mode of action related effect or safety of the drug) may be measured, based on newly emerging data from other ongoing studies and / or literature data.

Table 9-2: Sample types used for biomarker investigations

| Sample type, short form | Description |
|---|---|
| Biomarker serum | Blood sample for serum preparation for biomarker analysis |
| Biomarker plasma | Blood sample for plasma preparation for biomarker analysis |
| Biomarker urine | Urine sample for biomarker analysis |

# 9.4.3 Clinical efficacy variables

#### 9.4.3.1 Clinical outcome events

The following clinical outcome events will be collected:

- All deaths (CV and non-CV)
- HF hospitalizations and urgent visits for HF
- Myocardial infarction
- Stroke

The CEC will adjudicate all deaths as either CV or non-CV, and other events listed above in accordance with the pre-specified endpoint criteria in the adjudication charter. Investigators are mandated to report all suspected potential endpoints for adjudication by the CEC.

Events for adjudication should be reported as soon as critical data (as defined in the eCRF page) to the event adjudication is available. A query will be posted for events that require additional supporting documentation from the sites in order to render an adjudicated result and will be followed up by the sponsor. Every effort will be made to provide the CEC with clean eCRF data and required clinical data prior to event adjudication.

#### 9.4.3.2 NYHA class assessment

| NYHA<br>class | Symptoms |
|---|---|
| I | Patients with cardiac disease but without resulting limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea, or anginal pain. |
| II | Patients with cardiac disease resulting in slight limitation of physical activity. They are comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea, or anginal pain. |
| III | Patients with cardiac disease resulting in marked limitation of physical activity. They are comfortable at rest. Less than ordinary activity causes fatigue, palpitation, dyspnea, or anginal pain. |
| IV | Patients with cardiac disease resulting in inability to carry on any physical activity without discomfort. Symptoms of heart failure or the anginal syndrome may be present even at rest. If any physical activity is undertaken, discomfort is increased. |

Source: (45)




## 9.4.4 Patient-reported outcomes

At study visits where the questionnaire is required (see Table 9–1), patients should complete it before any other study procedures or assessments.

At collection, the questionnaire will be reviewed for completeness, and the patient will be encouraged to answer any blank data fields. Subsequently, a member of the investigator's team will enter the responses into the eCRF. Details about scoring and calculating algorithms will be provided in the SAP.

## 9.4.4.1 KCCQ

The **KCCQ** is the leading health-related quality-of-life measure for patients with CHF. It was developed in the late 1990s to early 2000s by Dr. John Spertus at the Mid-America Heart Institute, Kansas City, MO, USA. It is a 23-item questionnaire that independently measures the impact of patients' HF, or its treatment, on 7 distinct domains:

- 1) Symptom Frequency the KCCQ Symptom scale quantifies the frequency of clinical symptoms in HF, including fatigue, shortness of breath, paroxysmal nocturnal dyspnea, and edema / swelling.
- 2) Symptom Burden the KCCQ Symptom burden scale quantifies the severity of clinical symptoms in HF, including fatigue, shortness of breath and edema / swelling.
- 3) Physical Limitation the KCCQ Physical limitation scale measures the limitations patients experience, due to their HF, in performing routine activities.
- 4) Quality of Life the KCCQ Quality of life scale is designed to reflect patients' assessment of their quality of life, given the current status of their HF.
- 5) Social Limitations the KCCQ Social limitation scale quantifies the extent to which HF symptoms impair patients' abilities to interact in social roles.
- 6) Self-efficacy numerous studies have underscored the importance of patients being engaged in the management of their disease. The KCCQ Self-efficacy scale quantifies patients' perception of how to prevent HF exacerbations and manage complications when they arise.
- 7) Symptoms Stability—unlike the other 5 domains that provide cross-sectional quantification of patients' current status, the KCCQ Symptom stability domain measures recent changes in patients' symptoms. As a measure of change, it is most interpretable as a baseline assessment of the stability of patients' symptoms at the start of the study and thereafter.

In addition, there are 3 summary scores, a Total Symptom Score that combines the Symptom Frequency and the Symptom Burden scores, a Clinical Summary Score that combines the Total Symptom and Physical Limitation scores to replicate the NYHA classification; and an Overall Summary Score that includes the Total Symptom, Physical Limitation, Social Limitations, and Quality of Life scores (Figure 9–1).




Figure 9–1: KCCQ Scores



## 9.4.4.2 EQ-5D-5L

The EQ-5D-5L consists of 2 pages: the EQ-5D-5L descriptive system and the EQ visual analogue scale (EQ VAS). The EQ-5D-5L descriptive system comprises 5 dimensions: mobility, self-care, usual activities, pain / discomfort, and anxiety / depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The respondent is asked to indicate his / her health state by ticking (or placing a cross) in the box against the most appropriate statement in each of the 5 dimensions.

The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labeled 'the best health you can imagine' and 'the worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.

# 9.5 Pharmacokinetics / pharmacodynamics

It is planned to collect PK samples from all patients randomized. The data collected are intended to be used for PK analysis of the study population as a whole and should also give information about individual exposure to BAY 84-3174. Only the active metabolite BAY 84-3174 will be measured from the plasma samples collected (see Section 7.2 for details regarding different BAY numbers).

A sparse sampling schema has been developed, which will allow for a limited number of PK samples to be obtained from each patient. The sampling time points have been included in the flow chart (see Table 9–1). The PK sampling schedule is detailed in the visit description (Section 9.2). It is important to exactly record in the patient's file the time point when the PK sample is taken, as well as the times of the most recent medication intake prior to the blood sampling. The sampling variability will be used for modelling the PK and PD characteristics of the study medication.

Details about the collection, processing, storage and shipment of samples will be provided separately (e.g. sample handling sheets or laboratory manual).




# 9.6 Safety

## 9.6.1 Adverse events

#### 9.6.1.1 Definitions

## **Definition of adverse event (AE)**

In a clinical study, an AE is any untoward medical occurrence (i.e. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation subject after providing written informed consent for participation in the study. Therefore, an AE may or may not be temporally or causally associated with the use of a medicinal (investigational) product.

A surgical procedure that was planned prior to the start of the study by any physician treating the patient should not be recorded as an AE (however, the condition for which the surgery is required may be an AE).

In the following differentiation between medical history and AEs, the term "condition" may include abnormal physical examination findings, symptoms, diseases, laboratory, or ECG findings.

- Conditions that started before signing of informed consent and for which no symptoms
  or treatment are present until signing of informed consent are recorded as <u>medical</u>
  <u>history</u> (e.g. seasonal allergy without acute complaints).
- Conditions that started before signing of informed consent and for which symptoms or treatment are present after signing of informed consent, at unchanged intensity, are recorded as <a href="mailto:medical history">medical history</a> (e.g. allergic pollinosis).
- Conditions that started or deteriorated after signing of informed consent will be documented as adverse events.

### **Definition of serious adverse event (SAE)**

An SAE is classified as any untoward medical occurrence that, at any dose, meets any of the following criteria (a - f):

- a. Results in death
- b. Is life-threatening

The term 'life-threatening' in the definition refers to an event in which the patient was at risk of death at the time of the event, it does not refer to an event which hypothetically might have caused death if it were more severe.

c. Requires inpatient hospitalization or prolongation of existing hospitalization

A hospitalization or prolongation of hospitalization will not be regarded as an SAE if at least one of the following exceptions is met:

- The admission results in a hospital stay of less than 12 hours
- The admission is pre-planned




- -(e.g. elective or scheduled surgery arranged prior to the start of the study; admission is part of the study procedures as described in Section 9.2)
- The admission is not associated with an AE
   (e.g. social hospitalization for purposes of respite care).

However, it should be noted that invasive treatment during any hospitalization may fulfill the criterion of 'medically important' and as such may be reportable as an SAE dependent on clinical judgment. In addition, where local regulatory authorities specifically require a more stringent definition, the local regulation takes precedence.

- d. Results in persistent or significant disability / incapacity
  - Disability means a substantial disruption of a person's ability to conduct normal life's functions.
- e. Is a congenital anomaly / birth defect
- f. Is another serious or important medical event as judged by the investigator

### **Definition of treatment-emergent adverse event**

An AE is classified as treatment-emergent if it occurs or worsens after the first dose of study drug up to 6 weeks after the last dose of study drug.

### 9.6.1.2 Classifications for adverse event assessment

All AEs will be assessed and documented by the investigator according to the categories detailed below.

#### **9.6.1.2.1** Seriousness

For each AE, the seriousness must be determined according to the criteria given in Section 9.6.1.1

### 9.6.1.2.2 Intensity

The intensity of an AE is classified according to the following categories:

- Mild usually transient in nature and generally not interfering with normal activities
- Moderate sufficiently discomforting to interfere with normal activities
- Severe prevents normal activities

# 9.6.1.2.3 Causal relationship

The assessment of the causal relationship between an AE and the administration of treatment is a decision to be made by the investigator, who is a qualified physician, based on all information available at the time of the completion of the CRF.

The assessment is based on the question whether there was a "reasonable causal relationship" to the study treatment in question.

Possible answers are "yes" or "no".

An assessment of "no" would include:




1. The existence of a highly likely alternative explanation, e.g. mechanical bleeding at surgical site.

or

2. Non-plausibility, e.g. the patient is struck by an automobile when there is no indication that the drug caused disorientation that may have caused the event; cancer developing a few days after the first drug administration.

An assessment of "yes" indicates that that the AE is reasonably associated with the use of the study treatment.

Factors to be considered in assessing the relationship of the AE to study treatment include:

- The temporal sequence from drug administration: The event should occur after the drug is given. The length of time from drug exposure to event should be evaluated in the clinical context of the event.
- Recovery on drug discontinuation (de-challenge), recurrence on drug re-introduction (re-challenge): Patient's response after de-challenge or re-challenge should be considered in view of the usual clinical course of the event in question.
- Underlying, concomitant, intercurrent diseases:
   Each event should be evaluated in the context of the natural history and course of the disease being treated and any other disease the patient may have.
- Concomitant medication or treatment:
   The other drugs the patient is taking or the treatment the patient receives should be examined to determine whether any of them might have caused the event in question.
- Known response pattern for this class of drug.
- Exposure to physical and / or mental stresses: The exposure to stress might induce adverse changes in the recipient and provide a logical and better explanation for the event
- The pharmacology and pharmacokinetics of the study treatment:
   The pharmacokinetic properties (absorption, distribution, metabolism and excretion) of the study treatment, coupled with the individual patient's pharmacodynamics should be considered.
- The assessment is not possible.

#### Causal relationship to protocol-required procedure(s)

The assessment of a possible causal relationship between the AE and protocol-required procedure(s) is based on the question whether there was a "reasonable causal relationship" to protocol-required procedure(s).

Possible answers are "yes" or "no".




## 9.6.1.2.4 Action taken with study treatment

Any action on study treatment to resolve the AE is to be documented using the categories listed below.

- Drug withdrawn
- Drug interrupted
- Dose not changed
- Not applicable
- Unknown

# 9.6.1.2.5 Other specific treatment(s) of adverse events

- -None
- Remedial drug therapy
- -Other

#### 9.6.1.2.6 **Outcome**

The outcome of the AE is to be documented as follows:

- Recovered / resolved
- Recovering / resolving
- Recovered / resolved with sequelae
- Not recovered / not resolved
- Fatal
- Unknown

# 9.6.1.3 Assessments and documentation of adverse events

The investigator has to record on the respective CRF pages all adverse events occurring in the period between the signing of the informed consent and the end of the follow-up phase; after the end of the follow-up phase there is no requirement to actively collect AEs including deaths. The type of information that should be assessed and recorded by the investigator for each AE is listed in Section 9.6.1.2.

"Death" should not be recorded as an AE on the AE page. Instead, "death" is the outcome of an underlying AE(s).

For all serious adverse events (SAEs) the sponsor has to carry out a separate assessment for expectedness, seriousness and causal relationship to study drug.

### 9.6.1.4 Reporting of serious adverse events

The definition of serious adverse events (SAEs) is given in Section 9.6.1.1. Each SAE must be followed up until resolution or stabilization by submission of updated reports to the designated recipient.




If an SAE is unexpected, i.e. the event is not previously documented in the investigator's brochure (IB) (new occurrence) and is suspected to be related to the study drug, this event is considered a Suspected Unexpected Serious Adverse Reaction (SUSAR). In general, SUSARs will be unblinded by the sponsor for regulatory reporting (see below for exceptions).

### Investigator's notification of the sponsor

All investigators will be thoroughly instructed and trained on all relevant aspects of the investigator's reporting obligations for SAEs. This information, including all relevant contact details, is summarized in the investigator site file. This information will be updated as needed.

The investigator must report immediately (within 24 hours of the investigator's awareness) all SAEs occurring during the observation period defined in Section 9.6.1.3 to the recipient detailed in the instructions for SAE reporting included in the Investigator File. For this, an AE page and the complementary SAE pages in the CRF must be completed for each SAE.

SAEs occurring after the protocol-defined observation period will be processed by the sponsor according to all applicable regulations.

#### **Notification of the IECs/IRBs**

Notification of the IECs / IRBs about all relevant events (e.g. SAEs, SUSARs) will be performed by the sponsor and / or by the investigator according to all applicable regulations.

#### **Notification of the authorities**

The processing and reporting of all relevant events (e.g. SAEs, SUSARs) to the authorities will be done by the sponsor according to all applicable regulations.

# Sponsor's notification of the investigational site

The sponsor will inform all investigational sites about reported relevant events (e.g. SUSARs) according to all applicable regulations.

# Protocol-specific exceptions to SAE unblinding / reporting

If reported as SUSARs, the following clinical events will be exempted from unblinding and expedited reporting by the sponsor to investigators, IECs / IRBs, and regulatory agencies, since they are considered, consistent with the underlying condition, as disease related in the defined study population:

- CV death
- Worsening of heart failure
- Non-fatal myocardial infarction
- Non-fatal stroke
- Transient ischemic attack
- Cardiac arrhythmias
- Coronary revascularization procedures.




Note that all of these events will be reviewed and monitored by an external DMC unblinded to treatment as part of the overall assessment of safety and efficacy for neladenoson bialanate. Based upon their regular review of unblinded safety results, the DMC is empowered to make recommendations with regard to trial conduct to assure the continuing appropriate safety of the subjects participating in the study.

# 9.6.1.5 Expected adverse events

For this study, the applicable reference document is the most current version of the investigator's brochure (IB) for neladenoson bialanate.

Overview listings of frequent events that have occurred so far in the clinical development are shown in the current IB. If relevant new safety information is identified, the information will be integrated into an update of the IB and distributed to all participating sites.

The expectedness of AEs will be determined by the sponsor according to the applicable reference document and according to all local regulations.

# 9.6.1.6 Adverse events of special interest

Adverse events of special interest have to be reported to the sponsor along the timelines set for serious adverse events (even though they may not be classified as serious), i.e. within 24 hours of the investigator's awareness, as described in Section 9.6.1.4.

Adverse events of special interest are:

- Symptomatic bradycardia (HR < 50 bpm)
- Findings in ECG and / or AVIVO device as follows:
  - Mobitz type I AV-block leading to withdrawal or interruption of study drug
  - Mobitz type II AV block leading to withdrawal or interruption of study drug or leading to any change in therapy
  - o Third degree AV blocks

### 9.6.2 Pregnancies

Females of childbearing potential are excluded from the study. However, the investigator must report to the sponsor any pregnancy occurring in a female study patient during her participation in this study. The outcome of the pregnancy should be followed up carefully, and any outcome of the mother and the child at delivery should be reported.

The child's health should be evaluated at birth

For a pregnancy in the partner of a male study patient, all efforts will be made to obtain similar information on course and outcome, subject to the partner's consent.

For all reports, the forms provided are to be used. The investigator should submit them within the same timelines as an SAE.

# 9.6.3 Further safety

## 9.6.3.1 Laboratory evaluations

All laboratory evaluations will be done by central laboratory. Additional re-tests for liver monitoring (Section 9.6.3.6) will be done locally.




**Hematology:** erythrocytes, hemoglobin, hematocrit, MCV, MCH, MCHC, reticulocytes, leukocytes, differential blood count, platelets

Clinical chemistry: aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP), gamma glutamyl transpeptidase (GGT), lactate dehydrogenase (LDH), creatine kinase (CK), amylase, lipase, glucose, cholesterol (HDL, LDL, total), triglycerides, creatinine, urea, uric acid, bilirubin, total protein, albumin, sodium, potassium, calcium, chloride, magnesium, anorganic phosphate

**Coagulation:** partial thromboplastin time (PTT), international normalized ratio (INR)

# 9.6.3.2 Physical examination

The physical examination (by means of inspection, palpation, auscultation) will be performed by a physician at the investigational site covering at least the organs of the cardiovascular, respiratory, abdominal and neurological system.

Abnormal physical examination findings are recorded either as medical history or as adverse events (see Section 9.6.1.1).

### 9.6.3.3 12-lead ECG

The standard 12-lead ECG will be evaluated by the investigator and the following parameters will be recorded in the eCRF: HR, PR interval, QRSD interval, QT interval (uncorrected). QTcB (QT interval frequency-corrected according to Bazett's formula) will also be calculated but will not be valid for evaluation. The frequency-corrected QT interval will be calculated by data management according to the formulas of both Bazett and Fridericia.

All ECGs recorded during the study will be evaluated by a physician. He / she will document the diagnosis(es) including an overall assessment of the findings and their clinical relevance. Any clinically relevant abnormality will be documented as an AE or SAE.

# 9.6.3.4 Blood pressure and heart rate

Heart rate and blood pressure (systolic and diastolic) will be measured by a member of the investigator's study team with the patient at rest.

### 9.6.3.5 **AVIVO monitoring**

This section was changed in Amendment 2, see Section 15.1 for details.

AVIVO Mobile Patient Management System will be used to monitor patients' cardiovascular status as part of the safety assessment. The cardiac monitoring device will be worn as specified in Section 9.1.

The system is intended to continuously measure, record and periodically transmit ECG data. The system can detect (but is not limited to) higher degree AV-blocks > I°, SVTs (e.g. atrial fibrillation [AF], atrial flutter, paroxysmal SVTs), ventricular ectopy, bradyarrhythmias, conduction disorders and heart rate variability. Included in the service is the monitoring center - an independent certified diagnostic testing center staffed with ECG-trained technicians who read through the transmitted events 24h/7d. An electrophysiologist is also on staff for interpretation of difficult rhythms. The system has achieved CE mark and has US FDA clearance.




Apart from safety assessments, also the patient's everyday physical activity (e.g. duration, intensity) will be tracked.

Details of the cardiac monitoring and the device to be worn by the patient will be outlined in a manual that will be provided to all participating centers.

## 9.6.3.6 Liver function monitoring

Any patient with an ALT or AST > 3 x ULN or alkaline phosphatase (AP) >2 x ULN must be re-tested as soon as possible but at the latest within 48-72 hours of the investigator becoming aware of the result. This re-testing and any subsequent testing based on elevated levels should include measurement of ALT, AST, total and direct bilirubin, and AP, and will be assessed by local laboratory. Every effort should be made to clarify the etiology of elevated levels. Patient management is at the discretion of the investigator but the treating physician may continue the study drug during retesting. Liver function test monitoring should be performed as above for all patients even if the study drug is interrupted until tested values have normalized or returned to patient's baseline. If close liver monitoring is not possible then the patient should discontinue study medication.

For ALT or AST > 3 x ULN concurrent with a total bilirubin > 2 x ULN, every effort should be made to clarify any possible underlying disease(s).

The frequency of liver function tests based on re-test values is shown in Table 9–3.

Table 9-3: Liver function monitoring

| ALT, AST or AP level at re-test | Frequency | Further notice |
|---|---|---|
| ALT or AST > 3 x ULN | 2-3 times a week | Obtain details on liver related symptoms and exclude other causes of liver enzyme elevations |
| ALT or AST ≤ 3 x ULN | Once a week | Until return to normal or patient baseline levels |
| AP >2 x ULN | 2-3 times a week | Obtain details on liver related symptoms and exclude other causes of liver enzyme elevations |

Abbreviations: ALT = alanine aminotransferase; AP = alkaline phosphatase; AST = aspartate aminotransferase; ULN = upper limit of normal

Discontinuation of treatment should be considered if:

- ALT or AST > 8 x ULN
- ALT or AST > 5 x ULN for more than 2 weeks
- ALT or AST > 3 x ULN and (total bilirubin >2 x ULN or INR > 1.5)
- ALT or AST > 3 x ULN with the appearance of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash, and / or eosinophilia (> 5%)
- AP > 2 x ULN or ALT/AP < 2 for more than 2 weeks if other causes of cholestasis are excluded

## 9.7 Other procedures and variables

Not applicable.




# 9.8 Appropriateness of procedures / measurements

All parameters, as well as the methods to measure them, are standard variables / methods in clinical studies and / or clinical practice. They are widely used and generally recognized as reliable, accurate, and relevant.

# 10. Statistical methods and determination of sample size

### **10.1** General considerations

Statistical analyses will be performed by or under the supervision of the sponsor's study statistician and the assigned study statistical analyst using statistical analysis system (SAS); the version used will be specified in the statistical analysis plan (SAP).

A general description of the statistical methods to be used to analyze efficacy and safety in this is study is outlined below. A detailed SAP will be provided as a separate document that will be finalized and approved before database lock. The SAP will accommodate protocol amendments or unexpected issues in study execution or data that affect planned analyses and will provide more details on the analytical approaches, output tables and figures.

A meta-analysis of this study (15128) and of the study 17582 in patients with HFpEF, which is conducted at the same time, will be specified in a separate SAP.

# 10.2 Analysis sets

Documentation of protocol deviations and assignment of patients to analysis sets will be performed according to the sponsor's applicable Standard Operating Procedures and / or Operation Instructions.

The primary efficacy variables will be analyzed using the per-protocol set (PPS) and the full analysis set (FAS) for sensitivity analyses.

Data for all patients who signed informed consent but were not randomized will not be included in any statistical analyses except standard disposition tables and listings provided in the clinical study report (Screening failures and discontinued patients).

The statistical analysis sets are defined as follows:

#### **Full analysis set (FAS)**

The FAS population consists of all randomized unique patients. According to the ICH E9 guideline, this analysis set is as complete as possible and as close as possible to the intent-to-treat (ITT) ideal. Patients will be analyzed as randomized. The FAS will be used to display baseline characteristics and to display efficacy analyses.

### Safety analysis set (SAF)

The SAF population consists of all randomized patients who received at least one dose of study medication after randomization. The SAF will be used to display safety analyses. For safety analyses, patients will be analyzed as treated.




### **Per-protocol set (PPS)**

The PPS population consists of all FAS population patients without validity findings. Validity findings may include adherence and compliance issues and the violation of inclusion / exclusion criteria affecting efficacy evaluation. A list of potential validity findings will be provided in a separate protocol deviation document which will be finalized before database lock. The detailed definitions and the assignment of patients to this analysis set will be based on the validity review meeting. Patients will be analyzed as treated.

#### Pharmacokinetic analysis set (PKS)

The PKS population consists of all patients treated with neladenoson bialanate with at least 1 valid BAY 84-3174 plasma concentration and without protocol deviation that would interfere with the evaluation of the PK data.

# 10.3 Variables and planned statistical analyses

#### 10.3.1 Variables

### **10.3.1.1** Primary efficacy variables

- Absolute change from baseline in left ventricular ejection fraction (LVEF; %) after 20 weeks measured by echocardiography.
- Absolute change from baseline in log-transformed NT-proBNP (pg/mL) after 20 weeks, i.e., log-transformed NT-proBNP at Week 20 minus log-transformed NT-proBNP at baseline

# 10.3.1.2 Secondary efficacy variables

Secondary efficacy variables across different domains are:

- Key echocardiographic parameters, measured values and absolute change from baseline at 20 weeks:
  - o Left ventricular end-systolic volume (LVESV; mL)
  - o Left ventricular end-diastolic volume (LVEDV; mL)
- High sensitivity troponin T (hs-TNT; ng/L), measured values (log transformed) and absolute / relative change from baseline at 20 weeks as a biomarker of myocardial injury
- CV mortality, HF hospitalization and urgent visits for HF as clinical outcomes

## **10.3.1.3** Other exploratory variables

This section was changed in Amendment 2, see Section 15.1 for details.

- Activity (duration, intensity) reported values and absolute change from baseline at 20 weeks
- Echocardiographic parameters, as described in Section 9.4.1, measured values and absolute / relative change from baseline at 20 weeks
- Left ventricular ejection fraction (LVEF; %), measured values, number of patients in whom absolute change from baseline after 20 weeks is > 5%




- Mandatory biomarkers, as described in Section 9.4.2, measured values and absolute / relative change from baseline at 20 weeks, including
  - o NT-proBNP (pg/mL), measured values and relative change from baseline at 20 weeks to assess elevated filling pressures
  - o UACR, cystatin-C, NGAL for the evaluation of kidney function
- KCCQ and EQ-5D-5L, as described in Section 9.4.4, measured values and absolute / relative change from baseline
- All-cause mortality, non-fatal myocardial infarction, non-fatal stroke
- Change in NYHA class

### 10.3.1.4 Safety variables

Safety and tolerability variables are:

- Adverse events (Section 9.6.1), including
  - SAEs, AEs, treatment-emergent AEs and AEs of special interest, including AV blocks > I°
  - SAEs and AEs leading to discontinuation of interruption of study drug, including AV blocks in particular
- Laboratory abnormalities (Section 9.6.3.1), measured values and change from baseline, in particular
  - o Change in renal function measured by eGFR change from baseline
  - Change in liver function measured by bilirubin (total and fractions), AST and ALT from baseline
- 12-ECG abnormalities (Section 9.6.3.3) and PR interval duration
- Blood pressure and heart rate (Section 9.6.3.4); measured values and change from baseline
- Number of clinically significant findings in ECG and / or AVIVO device report

### 10.3.2 Statistical and analytical plans

All data will be listed and all variables will be summarized by means of descriptive statistics according to their type.

Summaries by treatment group using appropriate descriptive statistics will be provided for all study variables including demographic and baseline characteristics. Summary statistics will be presented for the original data as well as for the difference to baseline. Descriptive statistics such as arithmetic mean (or geometric mean, if applicable), median, standard deviation, quantiles, minimum, and maximum will be used to summarize continuous variables. Counts and percentages will be used to summarize categorical variables. Life tables and Kaplan-Meier estimates will be used to summarize time-to-event variables. Graphical data displays may also be used to summarize the data. Confidence intervals will be provided at a 2-sided level of 90% unless otherwise stated.

For this combined proof-of-concept and dose-finding study, an overall one-sided type I error level of 5% is planned to be used. The type I error will be controlled for the primary analysis of the primary variables.




There will be no formal control of the type I error for secondary or explorative analyses of the primary variables and any analysis of other efficacy variables.

# **10.3.2.1 Subgroups**

In order to assess the homogeneity of the dose response across the most important prognostic and predictive factors, subgroup analyses will be performed.

'Key' subgroups comprise:

- LVEF(%) at baseline: ≤25 vs. >25
- NT-proBNP (pg/ml) at baseline:  $\leq$  median vs. > median
- NYHA class at baseline: II vs. III / IV
- Prior β-blocker: yes vs. no

Truly exploratory analyses, i.e., mainly summary statistics, will be provided for a spectrum of demographic, disease and clinical characteristics, including

- Age (years): <65, 65-75, >75
- Gender: male vs. female
- Race: White vs. non-white
- Region: North America / South America / West Europe / East Europe / Asia
- Region: Japan vs. rest-of-the-world (analysis to be included in reports specific for Japan only)
- BMI at baseline (kg/m<sup>2</sup>):  $\leq$ 30 vs.  $\geq$ 30
- Time of CHF diagnosis to randomization (months):  $\leq 3$  vs.  $\geq 3$
- Prior hospitalization for heart failure: yes vs. no
- Etiology of CHF: ischemic vs. non-ischemic
- Diabetes: yes vs. no
- Atrial fibrillation: yes vs. no
- Hypertension: yes vs. no
- Prior CHF medication:
  - O Prior β-blocker in max tolerated dose: yes vs. no
  - o Prior use of ivabradine: yes vs. no
  - o Prior use of aldosterone antagonist: yes vs. no
  - o Prior use of ACE inhibitor: yes vs. no
  - o Prior use of ARB: yes vs. no
  - o Prior use of angiotensin receptor-neprilysin inhibitor (ARNI): yes vs. no
- Estimated GFR (ml/min/1.73 m<sup>2</sup>): <60 vs. >60

Further details will be described in detail in the SAP.




# 10.3.2.2 Analysis of the primary efficacy variables

This section was changed in Amendment 2, see Section 15.1 for details.

For both primary efficacy variables, it is planned to perform a test for a dose-response signal, respectively, under the assumption of a nearly monotone dose-response relationship in the dose range considered. The MCP-Mod method (46) combining multiple comparison procedures (MCP) principles with modeling techniques will be used for the primary statistical analysis of the primary efficacy variables. This method allows the flexibility of modeling for dose estimation, while preserving the robustness to model misspecification associated with MCP procedures.

Two primary variables have been defined to better evaluate multiple dimensions of the treatment effect, thereby adding a source of multiplicity. The overall outcome of the primary efficacy analysis will be considered positive if at least one of the two null hypotheses related to the primary efficacy variables can be rejected. The Hochberg (step-up) procedure will be applied to control the family-wise error rate (FWER):

Consider the null hypotheses for LVEF,  $H_{0,LVEF}$ , and for NT-proBNP,  $H_{0,NT\text{-proBNP}}$ , and their associated raw p-values  $p_{LVEF}$  and  $p_{NT\text{-proBNP}}$ . The Hochberg test is performed using the following steps:

- 1. If  $max(p_{LVEF}, p_{NT-proBNP}) \le \alpha = 0.05$ , both null hypotheses  $H_{0,LVEF}$  and  $H_{0,NT-proBNP}$  will be rejected and the procedure stops.
- 2. If  $\max(p_{\text{LVEF}}, p_{\text{NT-proBNP}}) > \alpha = 0.05$  and  $\min(p_{\text{LVEF}}, p_{\text{NT-proBNP}}) \le \alpha/2 = 0.025$ , the null hypothesis related to the larger p-value  $\max(p_{\text{LVEF}}, p_{\text{NT-proBNP}})$  will be accepted and the null hypothesis related to the smaller p-value  $\min(p_{\text{LVEF}}, p_{\text{NT-proBNP}})$  will be rejected.
- 3. Otherwise, both null hypotheses H<sub>0,LVEF</sub> and H<sub>0,NT-proBNP</sub> will be accepted.

# **Assumptions**

Five active doses of neladenoson bialanate will be used in this study: 5 mg, 10 mg, 20 mg, 30 mg, and 40 mg, as well as a placebo arm corresponding to a 0 mg dose.

The measurements of the primary efficacy variables are assumed to be normally distributed with the same standard deviation  $\sigma$  and independent between patients, respectively.

**LVEF**: The following assumptions were made for the absolute change from baseline in LVEF over 20 weeks:

- the expected mean effect under the placebo dose is conservatively assumed as an absolute increase from baseline of up to  $\Delta = 2\%$  with a standard deviation of  $\sigma = 7\%$
- while the maximum observable mean effect under neladenoson bialanate within the dose range considered is assumed as an absolute increase of  $\Delta = 5\%$  with a standard deviation of  $\sigma = 7\%$ .

This results in an expected maximum effect size of (5-2)/7 = 3/7 = 0.43 under conservative assumptions. Note that the threshold of clinical relevance is an absolute difference of 3% in the change from baseline over the placebo control group.




**NT-proBNP:** The following assumptions were made for the absolute change from baseline in the log-transformed NT-proBNP over 20 weeks:

- the expected mean effect under the placebo dose is assumed as an absolute decrease from baseline of -0.105 log(pg/mL) with a standard deviation of  $\sigma$  = 0.85 log(pg/mL), which is equivalent to a 10% relative reduction from a mean of 2,500 pg/mL at baseline.
- while the maximum observable mean effect under neladenoson bialanate within the dose range considered is assumed as an absolute decrease from baseline of -0.357 log(pg/mL) with a standard deviation of  $\sigma$  = 0.85 log(pg/mL), which is equivalent to a 30% relative reduction from a mean of 2,500 pg/mL at baseline.

It is assumed that the respective primary response efficacy variable, denoted as Y, is observed for the 6 parallel groups corresponding to doses levels: (placebo =)  $d_1 < d_2 < ... < d_k$ , where k = 6

For patient *j* within treatment group *i* the response can then be described by the following model:

$$Y_{ij} = f(d, \mathbf{\theta}) + \varepsilon_{ij}, \quad \varepsilon_{ij} \sim N(0, \sigma^2), \quad i = 1, ..., k, j = 1, ..., n_i,$$

where f(.) is parameterized by a vector of parameters  $\boldsymbol{\theta}$  and  $\varepsilon_{ij}$  is the error term.

A candidate set with M=5 different dose response shapes f(.) based on four models was chosen for the MCP-Mod method. Table 10–1 displays the response expressions for the shapes in the candidate sets for both, change in LVEF and change in log-transformed NT-proBNP. Figure 10–1 shows the corresponding dose-response shapes for change in LVEF. The model parameters were obtained through discussions with experts in the clinical team, taking prior beliefs and uncertainty into account. The dose-response shapes for NT-proBNP are equivalent to those for LVEF but with decreasing trends.

Table 10-1: Dose-response shapes used in the candidate set

| Model | Response as function of dose d | |
|---|---|---|
| | LVEF | NT-proBNP |
| Linear | 2 + 0.075 <i>d</i> | -0.105 - 0.0063d |
| Sigmoidal E <sub>max</sub> 1 | $2 + 3.007689d^4 / (9^4 + d^4)$ | -0.105 - 0.2526d4 / (94 + d4) |
| Sigmoidal E <sub>max</sub> 2 | $2 + 3.375d^3 / (20^3 + d^3)$ | -0.105 - 0.2835d3 / (203 + d3) |
| E <sub>max</sub> | 2 + 3.09375 <i>d</i> / (1.25 + <i>d</i> ) | -0.105 - 0.2599d / (1.25 + d) |
| Quadratic | $2 + 0.2d - 0.00333d^2$ | -0.105 - 0.0168d + 0.00028d <sup>2</sup> |




Model means (LVEF, absolute change from baseline in %) linear sigEmax1 sigEmax2 5 4 3 2 1 0 emax quadratic 10 20 30 40 Dose d in mg 4 3 2 1 20 30 0 30 0 10 40 10 20 40

Figure 10-1: Dose-response shapes used in the candidate set for change in LVEF

Abbreviations: LVEF = left ventricular ejection fraction

Based on the standardized versions of the models in the candidate set and the sample size allocation planned for this study, the optimum contrast coefficients for the 5 contrast tests on the dose-response shapes can be derived for both primary variables.

### **Analysis**

### Step 1: Detection of dose-response signal

For detecting an overall trend, or a dose-response signal, each of the M=5 dose-response shapes in the candidate set will be tested, using a single contrast test based on the updated version of contrast coefficients taking the actual sample sizes per treatment group into account.

For each model m, m = 1, ..., 5, in the candidate set

the null hypothesis

$$H_{0m}$$
:  $c_m \mu_m^0 = 0$ 

will be tested against

the respective 1-sided alternative hypothesis

$$H_{1m}: c_m \mu_m^0 > 0,$$

where 
$$\mu_m^0 = (\mu_{m1}^0, ..., \mu_{m6}^0)' = (f_m^0(d_1, \boldsymbol{\theta}_m^0), ..., f_m^0(d_6, \boldsymbol{\theta}_m^0))'$$
 and

 $f^0$  is the standardized version of the dose-response model  $f(d, \mathbf{\theta}) = \theta_0 + \theta_1 f^0(d, \mathbf{\theta}^0)$ . In this parameterization,  $\theta_0$  is a location parameter and  $\theta_1$  is a scale parameter such that only  $\mathbf{\theta}^0$  determines the shape of the model function.




A "proof-of-concept" dose-response relationship is detected if at least one single contrast test, is statistically significant, while controlling the family-wise error rate at level  $\alpha$ . The smallest of the corresponding adjusted p-values will be used for the Hochberg test.

This analysis will be performed for the FAS and PPS populations, where the PPS analysis is the primary analysis.

If no candidate model is statistically significant, the procedure stops, indicating that a dose-response relationship cannot be established from the observed data.

Out of the statistically significant models in the candidate set a best model can be selected for the next step: modeling and estimation.

### Step 2: Modeling and estimation of target doses

If a dose-response signal is established, the selected dose-response model(s) will be fitted to the observed data to estimate the model parameters.

The estimated dose-response model will be plotted against the doses including 90% confidence bands. Once the dose-response model has been successfully fitted to the data, target dose(s) of interest are estimated. Given a clinically relevant effect  $\Delta$ , a minimum effective dose  $(MED_{\Delta})$  associated with model  $f(d, \theta)$  is defined as

$$MED_{\Delta} = \operatorname{argmin}_{d \in (d_1, d_6]} \{ f(d, \mathbf{\theta}) \ge f(d_1, \mathbf{\theta}) + \Delta \}.$$

Estimates of  $MED_{\Delta}$  will be calculated for a clinically relevant change in LVEF assumed as  $\Delta = 3\%$  and potentially a plausible range of  $\Delta$  values which will be defined in the SAP. Estimation for change in log-transformed NT-proBNP will be performed analogously, ensuring an adequate back-transformation to allow for better interpretability of the results. In addition, estimates considering confidence bounds for the predicted value at a certain dose may be used. The final choice of the target dose depends on the evaluation of the primary efficacy variables and other efficacy variables, as well as safety considerations.

Modeling and estimation will be performed for the FAS and PPS populations as well as for relevant subgroups.

Further details will be described in the SAP.

As a secondary analysis pairwise comparisons of the active neladenoson bialanate dose groups with the placebo group will be performed without controlling the family-wise error rate.

## 10.3.2.3 Analysis of the secondary efficacy variables

The primary analysis of secondary efficacy variables will be performed in PPS, sensitivity analyses might be performed in the FAS. The secondary efficacy variables, except for the clinical outcomes, will be analyzed using similar statistical methods as for the primary efficacy variables, i.e. the MCP-Mod method with the same standardized candidate doseresponse shapes (with the proper direction: increasing or decreasing trend) and corresponding coefficients as for the primary variables. In addition to analyses comparing population means in the different dose groups, the number of patients in whom the individual change from baseline value crossed clinically meaningful thresholds will be analyzed. The totality of




evidence for the primary and secondary efficacy variables will be combined and used to assess the drug effect over dose levels.

Time to clinical outcome events since randomization (using both separate and composite outcomes) will be described by means of life table statistics and Kaplan-Meier estimates.

All other efficacy variables will be analyzed descriptively.

Further details will be described in the SAP.

## **10.3.2.4** Analysis of the safety variables

If not indicated otherwise, evaluation of safety variables will be done using the SAF.

#### **Adverse events**

The adverse events (AE) analysis will be performed as treated in the SAF. All tabulations will be descriptive only.

Individual listings of AEs will be provided. The incidence of treatment-emergent AEs and drug-related (treatment-emergent) AEs will be tabulated by treatment group using MedDRA terms. Separate tables and listing for serious AEs and death will be provided.

# **Further safety parameters**

The safety evaluation of laboratory data will include:

- Descriptive analysis of continuous laboratory parameters, and their changes from baseline by visit and treatment group.
- Incidence rates of treatment-emergent laboratory values outside of normal range by treatment group.
- Listings of laboratory data out of normal range.

Vital signs and their changes from baseline will be analyzed descriptively by visit and by treatment group.

ECG-findings (like AV-conduction abnormalities) will be summarized in frequency tables. A table displaying the number of patients with AV-block > I° will be provided.

Data from the AVIVO monitoring will be summarized; details will be described in the SAP.

Summary statistics and figures of heart rate and blood pressure (systolic, diastolic, and mean arterial pressure) will be created.

### 10.3.2.5 Pharmacokinetic analyses

Pharmacokinetic analyses will be performed on the population valid for pharmacokinetics.

For the investigation of systemic exposure to BAY 84-3174 and its relationship with treatment effects, the plasma concentrations of BAY 84-3174 will be determined at different time points using a sparse sampling approach in all participating patients (see Section 9.5). The plasma concentration vs. time data will be evaluated descriptively separated by dose and visit. Plots will be prepared pooling all individual plasma concentrations (naive pooling) vs. actual relative study times (time of sample collection after time of study drug administration).




Furthermore, the pharmacokinetic data and the relationship of markers of BAY 84-3174 exposure (e.g.  $C_{max}$ , AUC) with treatment effects will be evaluated using non-linear mixed effect modeling (NONMEM). The latter evaluation will be described in a separate analysis plan and will be reported under separate cover.

The PK bioanalysis will be performed under the responsibility of the Sponsor's Bioanalytics Laboratory.

# 10.3.2.6 Biomarker analyses

Biomarker data will be described by the following summary statistics: arithmetic mean, standard deviation, median, quantiles, minimum, and maximum.

Graphical displays of individual data as well as mean values with standard deviation will be included.

# 10.3.3 Missing data, censoring due to death, and drop outs

Generally, missing data will be handled as such, i.e., no imputation of missing data will be performed. An exception is the analysis of the primary and secondary efficacy variables (except for the clinical outcomes), as described below, and the timing of events relative to other events. For this purpose, data rules for the handling of missing or incomplete dates will be described in the SAP.

All missing or partial data will be presented in the patient data listing as they are recorded in the eCRF.

A number of descriptive analyses will be performed to better understand missing data patterns. The frequency, proportion and the reasons for premature discontinuation of both the study and study treatment will be reported. Kaplan-Meier plots for "time to end of study treatment (calculated as days from first dose to the earliest date of last dose, including premature stop of study medication and death)" and "time to end of study" will be provided, by treatment group and overall.

The number of patients who prematurely discontinue study participation or intake of study medication will be carefully evaluated with respect to the key baseline characteristics, which will be further specified in the SAP, and the reasons for premature discontinuation of study and / or study treatment. If the proportion of patients who withdraw across the dose groups is not fairly balanced, the impact on the primary variables will be further explored. To further explore the missingness pattern with regards to the "missing at random" assumption, the mean of the baseline values of the efficacy variable will be summarized for patients with and without post-baseline observations, by treatment group and overall.

For the analysis of the primary and secondary variables, it cannot necessarily be assumed that data are missing at random. As the choice of primary analysis will be based on assumptions that cannot be verified, the robustness of the results of the primary analysis will be investigated through appropriate sensitivity analyses making different assumptions, in accordance with the European Medicines Agency (EMA) "Guideline on missing data in confirmatory clinical trials".




## Efficacy analysis using the PPS

The primary efficacy analysis aims at evaluating the dose-response relationship of the primary and secondary efficacy variables (except for clinical outcomes) for all randomized patients who have remained in the study and adhered to study treatment according to the study protocol until Week 20 ("completers and treatment adherers" analysis). Therefore, the primary analysis will be performed in the per-protocol set, a subset of the FAS comprising "compliant and adherent" patients (as much as possible, defined via validity criteria). To avoid bias, the PPS will also include those "compliant and adherent" patients who are "censored" due to CV death or a hospitalization for HF preventing the assessment of the relevant efficacy endpoints 20 weeks after randomization to take place as planned. It is expected that these are the only patients for whom missing observations need to be considered in the primary analysis. A "worst case" approach will be used, where the missing change from baseline value will be imputed with a multiple of the worst change from baseline value, which is possible given the individual baseline value observed in the respective treatment group, or 0 if the worst change in that treatment group is positive for LVEF / negative for NT-proBNP.

As a sensitivity analysis, a "completers and treatment adherers" only analysis excluding the censored patients in the per-protocol analysis set will be performed. This strategy leads to unbiased estimates only if missing values are "missing completely at random" (MCAR), i.e. the missingness – including missing data due to death – is independent of both observed and unobserved outcomes. This condition is unlikely to hold exactly but rather approximately.

Further sensitivity analyses on the PPS may be performed if the missing data patterns suggest further exploration.

# Efficacy analysis using the FAS

The efficacy analysis in the FAS aims at evaluating the dose-response relationship of the primary and secondary efficacy variables for all randomized patients. Efficacy analyses in the FAS will include the following:

- Generally, it will be assumed that missing observations for the respective efficacy variables are missing at random. This implies that the behavior of the post dropout observations can be predicted from the observed variables using appropriate imputation models. Likely exceptions to the missing at random assumption are observations which are missing due to a patient's CV death or HF hospitalization prior to the visit in Week 20. These observations can be assumed to be missing not at random (MNAR), i.e., that missingness depends both on observed and unobserved outcomes and that an explicit model for the patient's statistical behavior after drop-out (or death) is required. Therefore, an analysis based on a pattern mixture framework (47) with different imputation rules depending on the reason for missingness will be used using a multiple imputation model, followed by a modification of the imputed data applying penalties:
  - 1. First, multiple imputation will be applied to draw sets of completed data, using an appropriate imputation model. Baseline characteristics which should be considered in the imputation model include but are not restricted to the baseline values of the respective efficacy variable, the treatment group, and sex.




- 2. The imputed data will be modified by applying penalties. The choice of the penalty may be guided by the worst observed change from baseline for the respective outcome in the corresponding treatment group, e.g. by choosing the penalty as a multiple of the worst observed change from baseline value.
- 3. After modifying the completed data sets, the primary analysis using the MCP-step of the MCP-Mod methodology will be applied to the multiply imputed datasets and the results will be combined.
- An analysis where for each patient without an observation at the visit in Week 20 the missing value will be imputed according to a last observation carried forward approach, including the baseline value. Such an analysis is usually biased but will make use of the observations obtained at early EOT visits.

For reproducibility, the SAS seed number for creating the random numbers for the multiple imputation will be set to the study number. More details will be described in the SAP.

# **10.4** Determination of sample size

In the first step, this combined proof-of-concept and Phase IIb dose-finding study has been powered for the detection of a dose response signal in the primary efficacy variable change in LVEF.

The sample size for the primary efficacy variable change in LVEF was evaluated under the assumptions described in Section 10.3.2.2 and a type I error level = 5% with the aim to achieve at least 80% power for the one-sided primary multiple contrast test. The overall randomization ratio was assumed to be 3:1:2:2:2:2 for doses 0, 5, 10, 20, 30, and 40 mg.

Table 10–2 displays the power for the multiple contrast test in the MCP-Mod approach, used as primary analysis, for the set of specified alternatives.

| Sample size | | Power for alternative based on respective dose-response model (in %) | | | | | |
|---|---|---|---|---|---|---|---|
| Overall | Per | Linear | Sigmoidal | Sigmoidal | $E_{max}$ | Quadratic | Minimum |
| | group <sup>a</sup> | | E <sub>max</sub> 1 | E <sub>max</sub> 2 | | | |
| 240 | 40 | 73.36 | 86.24 | 81.20 | 82.26 | 79.97 | 73.36 |
| 252 | 42 | 75.26 | 87.73 | 82.94 | 83.94 | 81.70 | 75.26 |
| 264 | 44 | 77.10 | 89.13 | 84.58 | 85.58 | 83.31 | 77.10 |
| 276 | 46 | 78.71 | 90.30 | 85.97 | 86.94 | 84.70 | 78.71 |
| 288 | 48 | 80.31 | 91.39 | 87.30 | 88.25 | 86.09 | 80.31 |
| 300 | 50 | 81.62 | 92.27 | 88.42 | 89.32 | 87.24 | 81.62 |
| 312 | 52 | 82.99 | 93.15 | 89.53 | 90.38 | 88.39 | 82.99 |
| 324 | 54 | 84.25 | 93.92 | 90.54 | 91.37 | 89.50 | 84.25 |
| 336 | 56 | 85.43 | 94.60 | 91.45 | 92.22 | 90.39 | 85.43 |
| 348 | 58 | 86.56 | 95.22 | 92.31 | 93.02 | 91.28 | 86.56 |

Table 10-2: Power for multiple contrast test for set of different alternatives

To achieve at least 80% power for the multiple contrast test in the MCP-Mod approach under all different alternatives, a minimum of 48 patients per treatment group (72 patients for the placebo and 24 patients for the 5 mg group) is needed, resulting in an overall sample size of N = 288 patients.

A Number of patients randomized to dose levels 10 mg, 20 mg, 30 mg, and 40 mg of neladenoson bialanate, for placebo sample size per group to be multiplied by 3/2, for dose level 5 mg sample size per group to be divided by 2.




In the second step, the power for the multiple contrast test in the MCP-Mod approach for the absolute change in log-transformed NT-proBNP was estimated, based on the assumptions outlined in Section 10.3.2.2 and a given sample size of N = 288. Statistical simulations were used to assess the power of the Hochberg test to reject at least one of the two null hypotheses. It was concluded that an overall sample size of N = 288 patients is sufficient to reject at least one of the two primary efficacy hypotheses with a power of about 83%.

This power would drop to less than 80%, if the relative reduction of NT-proBNP from baseline within the investigated dose range for neladenoson bialanate is < 27.5% compared to an expected reduction from baseline of 10% under placebo.

Based on these considerations, a total of 384 patients are planned to be randomized to the 6 treatment groups:

- 96 patients are planned to be randomized to placebo (0 mg),
- 64 patients each are planned to be randomized to the dose levels 10 mg, 20 mg, 30 mg, and 40 mg of neladenoson bialanate, and
- 32 patients are planned to be randomized to the dose level 5 mg of neladenoson bialanate.

These numbers already include adequate assumptions on expected drop-out after randomization and invalid or missing data. In the selected population it is expected that only about 75% of all randomized patients, i.e. about 288 patients, will contribute complete data to the primary analysis in the PPS.

All power estimations and simulations were performed with the DoseFinding package in R, version 3.0.2 (2013-09-25).

### 10.5 Planned interim analyses

A formal interim analysis is not planned. Periodic data review by a DMC will be performed to monitor safety.

# 11. Data handling and quality assurance

## 11.1 Data recording

This section was changed in Amendment 2, see Section 15.1 for details.

The data collection tool for this study will be a validated electronic data capture system called RAVE. Patient data necessary for analysis and reporting will be entered / transmitted into a validated database or data system (e.g. TOSCA; SAS).

Data required according to this protocol will be recorded by investigational site personnel via data entry into the internet based EDC software system RAVE, which Bayer has licensed from Medidata Solutions Worldwide. RAVE has been validated by Medidata Solutions Worldwide and Bayer for use in its clinical studies. RAVE allows for the application of software logic to set-up data entry screens and data checks to ensure the completeness and accuracy of the data entered by the site personnel. Bayer extensively applies the logic to ensure data are complete and reflect the clinical data requirements of the study. Data queries

## Integrated Clinical Study Protocol No. BAY 1067197 / 15128




resulting from the application of the software logic are resolved by the site personnel. The data are stored at a secure host facility maintained by Medidata Solutions Worldwide and transferred on a periodic basis to Bayer's internal computer system via a secure Virtual Private Network.

All access to the RAVE system is through a password-protected security system that is part of the RAVE software. All internal Bayer and external investigator site personnel seeking access must go through a thorough RAVE training process before they are granted access to RAVE for use in Bayer's clinical studies. Training records are maintained.

All personnel with access to the RAVE system are supported by a Service Desk staffed with trained personnel to answer questions and ensure access is maintained such that data entry can proceed in a timely manner.

The RAVE System contains a system-generated audit trail that captures any changes made to a data field, including who made the change, why the change was made and the date and time it was made. This information is available both at the investigator's site and at Bayer. Data entries made in the RAVE EDC screens are supported by source documents maintained for all patients enrolled in this study.

#### **Source documentation**

The site must implement processes to ensure availability of all required source documentation. A source document checklist (not part of this protocol) will be used at the site to identify the source data for key data points collected and the monitor will work with the site to complete this.

It is the expectation of the sponsor that all data entered into the CRF has source documentation available at the site.

#### Data recorded from screening failures

At minimum, the following data should be recorded in the CRF:

- Demographic information (patient number; year of birth / age; sex; if permitted locally, race / ethnicity)
- Date of informed consent
- Inclusion / exclusion criteria
- Reason for premature discontinuation
  - o AE information, if applicable
- Date of last visit.

These data will be transferred to the respective database.

For screening failures with an SAE, the following data should be collected in the CRF in addition to the data specified above:




- All information related to the SAE such as:
  - The SAE itself
  - Concomitant medication
  - Medical history
  - Other information needed for SAE complementary page

# 11.2 Monitoring

In accordance with applicable regulations, GCP, and sponsor's / CRO's procedures, monitors will contact the site prior to the start of the study to review with the site staff the protocol, study requirements, and their responsibilities to satisfy regulatory, ethical, and sponsor's requirements. When reviewing data collection procedures, the discussion will also include identification and documentation of source data items.

The sponsor / designee will monitor the site activity to verify that the:

- Data are authentic, accurate and complete. Supporting data may be requested (example: blood glucose readings to support a diagnosis of diabetes).
- Safety and rights of patients are being protected
- Study is conducted in accordance with the currently approved protocol (including study treatment being used in accordance with the protocol)
- Any other study agreements, GCP, and all applicable regulatory requirements are met.

The investigator and the head of the medical institution (where applicable) agrees to allow the monitor direct access to all relevant documents.

# 11.3 Data processing

Data will be collected as described in Section 11.1. Clinical data management will be performed in accordance with sponsor's applicable standards and data cleaning procedures. This is applicable for data recorded in the eCRF as well as for data from other sources (e.g. IxRS, laboratory, ECG, AVIVO).

For data coding (e.g. AEs, medication), internationally recognized and accepted dictionaries will be used.

After its initial release for biometrical analysis, the clinical database is planned to be reopened for the inclusion of the following additional data: pharmacokinetic data and biomarker data.

## 11.4 Missing data

The following measures will be implemented to minimize the amount of missing data.

• Encourage further participation in the study, i.e. phone call 26 weeks after the start of treatment, even if the study medication is discontinued early.




- If the patient does not attend the visits in person, the investigator should make every effort to collect information on mortality and / or hospitalization from other sources, e.g. family / friend / general physician / etc.
- Ask sites to call patients the day before certain study visits to remind them to remember
  the time they take their study medication and to remind them in case study medication
  should not be taken at home the next day.
- Educate patients on the AVIVO device and train sites to prepare the patient's skin for adherence of the sensor. Ask sites to call patients at the end of the wearing period to provide instructions for removal, storage and return at the next visit.
- Try to avoid unnecessary patient withdrawals (see Section 6.4).

### 11.5 Audit and inspection

To ensure compliance with GCP and regulatory requirements, a member of the sponsor's (or a designated CRO's) quality assurance unit may arrange to conduct an audit to assess the performance of the study at the study site and of the study documents originating there. The investigator / institution will be informed of the audit outcome.

In addition, inspections by regulatory health authority representatives and IEC(s) / IRB(s) are possible. The investigator should notify the sponsor immediately of any such inspection.

The investigator / institution agrees to allow the auditor or inspector direct access to all relevant documents and allocate his / her time and the time of his / her staff to the auditor / inspector to discuss findings and any issues. Audits and inspections may occur at any time during or after completion of the study.

# 11.6 Archiving

Essential documents shall be archived safely and securely in such a way that ensures that they are readily available upon authorities' request.

Patient (hospital) files will be archived according to local regulations and in accordance with the maximum period of time permitted by the hospital, institution or private practice. Where the archiving procedures do not meet the minimum timelines required by the sponsor (minimum is 25 years; longer if required by local regulation), alternative arrangements must be made to ensure the availability of the source documents for the required period.

The investigator / institution notifies the sponsor if the archival arrangements change (e.g. relocation or transfer of ownership).

The investigator site file is not to be destroyed without the sponsor's approval.

The contract with the investigator / institution will contain reference to all regulations relevant for the study center.




# 12. Premature termination of the study

The sponsor has the right to close this study (or, if applicable, individual segments thereof [e.g. treatment arms; dose steps; centers]) at any time, which may be due but not limited to the following reasons:

- If risk-benefit ratio becomes unacceptable owing to, for example,
  - Safety findings from this study (e.g. SAEs)
  - Results of parallel clinical studies
  - Results of parallel animal studies (on e.g. toxicity, teratogenicity, carcinogenicity or reproduction toxicity).
- If the study conduct (e.g. recruitment rate; drop-out rate; data quality; protocol compliance) does not suggest a proper completion of the trial within a reasonable time frame.

The investigator has the right to close his / her center at any time.

For any of the above closures, the following applies:

- Closures should occur only after consultation between involved parties. Final decision on the closure must be in writing.
- All affected institutions (e.g. IEC(s) / IRB(s); competent authority(ies); study center; head of study center) must be informed as applicable according to local law.
- All study materials (except documentation that has to remain stored at site) must be returned to the sponsor. The investigator will retain all other documents until notification is given by the sponsor for destruction.
- In the event of a partial study closure, ongoing patients, including those in post study follow-up, must be taken care of in an ethical manner.

Details for individual patient's withdrawal can be found in Section 6.4.1.

# 13. Ethical and legal aspects

# 13.1 Investigator(s) and other study personnel

This section was changed in Amendment 2, see Section 15.1 for details.

Sponsor's study medical expert is identified on the Title page.

Coordinating investigators in this study will be:








All other study personnel not included in this section are identified in a separate personnel list (not part of this clinical study protocol) as appropriate. This list will be updated as needed; an abbreviated version with personnel relevant for the centers will be available in each center's investigator site file.

Whenever the term 'investigator' is noted in the protocol text, it may refer to either the principal investigator at the site, or an appropriately qualified, trained and delegated individual of the investigational site.

The principal investigator of each center must sign the protocol signature page and must receive all required external approvals (e.g. health authority, ethics committee, sponsor) before patient recruitment may start at the respective center. Likewise, all amendments to the protocol must be signed by the principal investigator and must receive all required external approvals before coming into effect at the respective center.

A complete list of all participating centers and their investigators, as well as all required signature documents, will be maintained in the sponsor's study file.

The global sponsor of this study is identified on the title page of this protocol. If required by local law, local co-sponsors will be nominated; they will be identified on the respective country-specific signature pages.

#### External data evaluation bodies

### **Steering Committee**

The main task of the Steering Committee, which is composed of a panel of experts in the field, is to support the conduct of the study and to advise the sponsor on clinical, medical, and scientific questions. Details of the committee will be specified in the Steering Committee charter.

### **Data Monitoring Committee**

Ongoing safety monitoring during the conduct of the study will be performed by an external and unblinded DMC. Analysis periods and procedures will be defined in an operational charter (DMC Charter) filed in the study file. Following data review, the DMC will provide written recommendations that will be transferred to Bayer. All other definitions will be provided in the DMC charter.




#### **Clinical Events Committee**

Blinded adjudication of all hospitalizations, urgent visits for HF and deaths will be performed by a central CEC as described in the CEC charter. Data entry procedures and documentation necessary for case adjudication will also be described in the CEC charter. Adjudication results will be the basis for the final analysis.

# 13.2 Funding and financial disclosure

### **Funding**

This study will be funded by its sponsor.

#### Financial disclosure

Each investigator (including principal and / or any sub investigators) who is directly involved in the treatment or evaluation of research patients has to provide a financial disclosure according to all applicable legal requirements. All relevant documentation will be filed in the trial master file.

# 13.3 Ethical and legal conduct of the study

The procedures set out in this protocol, pertaining to the conduct, evaluation, and documentation of this study, are designed to ensure that the sponsor and investigator abide by Good Clinical Practice (GCP) guidelines and the guiding principles detailed in the Declaration of Helsinki. The study will also be carried out in keeping with applicable local law(s) and regulation(s).

Documented approval from appropriate IEC(s) / IRBs will be obtained for all participating centers / countries before start of the study, according to GCP, local laws, regulations and organizations. When necessary, an extension, amendment or renewal of the IEC / IRB approval must be obtained and also forwarded to the sponsor. The responsible unit (e.g. IEC / IRB, head of the study center / medical institution) must supply to the sponsor, upon request, a list of the EC / IRB members involved in the vote and a statement to confirm that the IEC / IRB is organized and operates according to GCP and applicable laws and regulations.

Strict adherence to all specifications laid down in this protocol is required for all aspects of study conduct; the investigator may not modify or alter the procedures described in this protocol.

Modifications to the study protocol will not be implemented by either the sponsor or the investigator without agreement by both parties. However, the investigator or the sponsor may implement a deviation from, or a change of, the protocol to eliminate an immediate hazard(s) to the trial subjects without prior IEC / IRB / sponsor approval / favorable opinion. As soon as possible, the implemented deviation or change, the reasons for it and if appropriate the proposed protocol amendment should be submitted to the IEC / IRB / head of medical institution / sponsor. Any deviations from the protocol must be explained and documented by the investigator.

Details on discontinuation of the entire study or parts thereof can be found in Section 12.



#### 13.4 Patient information and consent

All relevant information on the study will be summarized in an integrated patient information sheet and informed consent form provided by the sponsor or the study center. A sample patient information and informed consent form is provided as a document separate to this protocol.

Based on this patient information sheet, the investigator or designee will explain all relevant aspects of the study to each patient prior to his / her entry into the study (i.e. before any examinations and procedures associated with the selection for the study are performed or any study-specific data is recorded on study-specific forms).

The investigator will also mention that written approval of the IRB / IEC has been obtained.

Each patient will be informed about the following aspects of premature withdrawal:

- Each patient has the right to withdraw from the study at any time without any disadvantage and without having to provide reasons for this decision.
- The patient's consent covers end-of-study examinations as specified in the visit description described in Section 9.2 to be conducted after withdrawal of consent to treatment.
- The patient's data that have been collected until the time of withdrawal will be retained and statistically analyzed in accordance with the statistical analysis plan.
- Patient-specific data on the basis of material obtained before withdrawal may be generated after withdrawal (e.g. image reading, analysis of biological specimen such as blood, urine or tissues); these data would also be retained and statistically analyzed in accordance with the statistical analysis plan. The patient has the right to object to the generation and processing of this post-withdrawal data. The patient's oral objection may be documented in the patient's source data.

Each patient will have ample time and opportunity to ask questions.

Only if the patient voluntarily agrees to sign the informed consent form and has done so, may he / she enter the study. Additionally, the investigator will personally sign and date the form. The patient will receive a copy of the signed and dated form.

The signed informed consent statement is to remain in the investigator site file or, if locally required, in the patient's note / file of the medical institution.

In the event that informed consent is obtained on the date that baseline study procedures are performed, the study record or patient's clinical record must clearly show that informed consent was obtained prior to these procedures.

The informed consent form and any other written information provided to patients will be revised whenever important new information becomes available that may be relevant to the patient's consent, or there is an amendment to the protocol that necessitates a change to the content of the patient information and / or the written informed consent form. The investigator will inform the patient of changes in a timely manner and will ask the patient to confirm his/her participation in the study by signing the revised informed consent form. Any revised written informed consent form and written information must receive the IEC / IRB's approval / favorable opinion in advance of use.




## 13.5 Publication policy and use of data

The sponsor has made the information regarding the study protocol publicly available on the internet at www.clinicaltrials.gov.

All data and results and all intellectual property rights in the data and results derived from the study will be the property of the sponsor who may utilize them in various ways, such as for submission to government regulatory authorities or disclosure to other investigators.

Regarding public disclosure of study results, the sponsor will fulfill its obligations according to all applicable laws and regulations. The sponsor is interested in the publication of the results of every study it performs.

The sponsor recognizes the right of the investigator to publish the results upon completion of the study. However, the investigator, whilst free to utilize study data derived from his / her center for scientific purposes, must obtain written consent of the sponsor on the intended publication manuscript before its submission. To this end, the investigator must send a draft of the publication manuscript to the sponsor within a time period specified in the contract. The sponsor will review the manuscript promptly and will discuss its content with the investigator to reach a mutually agreeable final manuscript.

## 13.6 Compensation for health damage of patients / insurance

The sponsor maintains clinical trial insurance coverage for this study in accordance with the laws and regulations of the country in which the study is performed.

## 13.7 Confidentiality

All records identifying the patient will be kept confidential and, to the extent permitted by the applicable laws and / or regulations, will not be made publicly available.

Patient names will not be supplied to the sponsor. Only the patient number will be recorded in the CRF, and if the patient name appears on any other document (e.g. pathologist report), it must be obliterated before a copy of the document is supplied to the sponsor. Study findings stored on a computer will be stored in accordance with local data protection laws. As part of the informed consent process, the patients will be informed in writing that representatives of the sponsor, IEC / IRB, or regulatory authorities may inspect their medical records to verify the information collected, and that all personal information made available for inspection will be handled in strictest confidence and in accordance with local data protection laws.

If the results of the study are published, the patient's identity will remain confidential.

The investigator will maintain a list to enable patients to be identified.




## 14. Reference list

- 1. McMurray JJ, Adamopoulos S, Anker SD, Auricchio A, Bohm M, Dickstein K, et al. ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure 2012: The Task Force for the Diagnosis and Treatment of Acute and Chronic Heart Failure 2012 of the European Society of Cardiology. Developed in collaboration with the Heart Failure Association (HFA) of the ESC. Eur Heart J. 2012;33(14):1787-847.
- 2. Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Blaha MJ, et al. Heart disease and stroke statistics--2014 update: a report from the American Heart Association. Circulation. 2014;129(3):e28-e292.
- 3. Mosterd A, Hoes AW. Clinical epidemiology of heart failure. Heart. 2007;93(9):1137-46.
- 4. McCullough PA, Philbin EF, Spertus JA, Kaatz S, Sandberg KR, Weaver WD, et al. Confirmation of a heart failure epidemic: findings from the Resource Utilization Among Congestive Heart Failure (REACH) study. Journal of the American College of Cardiology. 2002;39(1):60-9.
- 5. Stewart S, MacIntyre K, Hole DJ, Capewell S, McMurray JJ. More 'malignant' than cancer? Five-year survival following a first admission for heart failure. European journal of heart failure. 2001;3(3):315-22.
- 6. Executive summary: HFSA 2006 Comprehensive Heart Failure Practice Guideline. J Card Fail. 2006;12(1):10-38.
- 7. Gheorghiade M, Vaduganathan M, Fonarow GC, Bonow RO. Rehospitalization for heart failure: problems and perspectives. Journal of the American College of Cardiology. 2013;61(4):391-403.
- 8. SOLVD. Effect of enalapril on survival in patients with reduced left ventricular ejection fractions and congestive heart failure. The SOLVD Investigators. N Engl J Med. 1991;325(5):293-302.
- 9. Packer M, Bristow MR, Cohn JN, Colucci WS, Fowler MB, Gilbert EM, et al. The effect of carvedilol on morbidity and mortality in patients with chronic heart failure. U.S. Carvedilol Heart Failure Study Group. N Engl J Med. 1996;334(21):1349-55.
- Pitt B, Zannad F, Remme WJ, Cody R, Castaigne A, Perez A, et al. The effect of spironolactone on morbidity and mortality in patients with severe heart failure. Randomized Aldactone Evaluation Study Investigators. N Engl J Med. 1999;341(10):709-17.
- 11. McMurray JJ, Packer M, Desai AS, Gong J, Lefkowitz MP, Rizkala AR, et al. Angiotensin-neprilysin inhibition versus enalapril in heart failure. N Engl J Med. 2014;371(11):993-1004.
- 12. Gheorghiade M, Bohm M, Greene SJ, Fonarow GC, Lewis EF, Zannad F, et al. Effect of aliskiren on postdischarge mortality and heart failure readmissions among patients hospitalized for heart failure: the ASTRONAUT randomized trial. Jama. 2013;309(11):1125-35.




- 13. Gheorghiade M, Greene SJ, Filippatos G, Erdmann E, Ferrari R, Levy PD, et al. Cinaciguat, a soluble guanylate cyclase activator: results from the randomized, controlled, phase IIb COMPOSE programme in acute heart failure syndromes. Eur J Heart Fail. 2012;14(9):1056-66.
- 14. Bayeva M, Gheorghiade M, Ardehali H. Mitochondria as a therapeutic target in heart failure. Journal of the American College of Cardiology. 2013;61(6):599-610.
- 15. Sabbah HN, Gupta RC, Kohli S, Wang M, Rastogi S, Zhang K, et al. Chronic therapy with a partial adenosine A1-receptor agonist improves left ventricular function and remodeling in dogs with advanced heart failure. Circulation Heart failure. 2013;6(3):563-71.
- 16. Sabbah HN, Sharov V, Riddle JM, Kono T, Lesch M, Goldstein S. Mitochondrial abnormalities in myocardium of dogs with chronic heart failure. J Mol Cell Cardiol. 1992;24(11):1333-47.
- 17. Sharov VG, Goussev A, Lesch M, Goldstein S, Sabbah HN. Abnormal mitochondrial function in myocardium of dogs with chronic heart failure. J Mol Cell Cardiol. 1998;30(9):1757-62.
- 18. Sharov VG, Todor AV, Silverman N, Goldstein S, Sabbah HN. Abnormal mitochondrial respiration in failed human myocardium. J Mol Cell Cardiol. 2000;32(12):2361-7.
- 19. Sharov VG, Todor A, Khanal S, Imai M, Sabbah HN. Cyclosporine A attenuates mitochondrial permeability transition and improves mitochondrial respiratory function in cardiomyocytes isolated from dogs with heart failure. J Mol Cell Cardiol. 2007;42(1):150-8.
- 20. Neubauer S. The failing heart--an engine out of fuel. N Engl J Med. 2007;356(11):1140-51.
- 21. Hasenfuss G, Pieske B. Calcium cycling in congestive heart failure. J Mol Cell Cardiol. 2002;34(8):951-69.
- 22. Conraads VM, Van Craenenbroeck EM, De Maeyer C, Van Berendoncks AM, Beckers PJ, Vrints CJ. Unraveling new mechanisms of exercise intolerance in chronic heart failure: role of exercise training. Heart Fail Rev. 2013;18(1):65-77.
- 23. Nell PG, Albrecht-Kupper B. The adenosine A1 receptor and its ligands. Prog Med Chem. 2009;47:163-201.
- 24. Hwang SJ, Melenovsky V, Borlaug BA. Implications of coronary artery disease in heart failure with preserved ejection fraction. Journal of the American College of Cardiology. 2014;63(25 Pt A):2817-27.
- 25. Rusinaru D, Houpe D, Szymanski C, Levy F, Marechaux S, Tribouilloy C. Coronary artery disease and 10-year outcome after hospital admission for heart failure with preserved and with reduced ejection fraction. European journal of heart failure. 2014;16(9):967-76.
- 26. Baxter GF, Hale SL, Miki T, Kloner RA, Cohen MV, Downey JM, et al. Adenosine A1 agonist at reperfusion trial (AART): results of a three-center, blinded, randomized, controlled experimental infarct study. Cardiovascular drugs and therapy / sponsored by the International Society of Cardiovascular Pharmacotherapy. 2000;14(6):607-14.




- 27. Veres G, Radovits T, Otila G, Hirschberg K, Haider H, Krieger N, et al. Efficacy of the non-adenosine analogue A1 adenosine receptor agonist (BR-4935) on cardiovascular function after cardiopulmonary bypass. The Thoracic and cardiovascular surgeon. 2010;58(2):86-92.
- 28. Bott-Flugel L, Bernshausen A, Schneider H, Luppa P, Zimmermann K, Albrecht-Kupper B, et al. Selective attenuation of norepinephrine release and stress-induced heart rate increase by partial adenosine A1 agonism. PloS one. 2011;6(3):e18048.
- 29. Richardt G, Waas W, Kranzhofer R, Mayer E, Schomig A. Adenosine inhibits exocytotic release of endogenous noradrenaline in rat heart: a protective mechanism in early myocardial ischemia. Circ Res. 1987;61(1):117-23.
- 30. Cavender MA, Steg PG, Smith SC, Eagle K, Ohman EM, Goto S, et al. Impact of Diabetes on Hospitalization for Heart Failure, Cardiovascular Events, and Death: Outcomes at 4 Years from the REACH Registry. Circulation. 2015.
- 31. Fredholm BB, AP IJ, Jacobson KA, Klotz KN, Linden J. International Union of Pharmacology. XXV. Nomenclature and classification of adenosine receptors. Pharmacol Rev. 2001;53(4):527-52.
- 32. Massie BM, O'Connor CM, Metra M, Ponikowski P, Teerlink JR, Cotter G, et al. Rolofylline, an adenosine A1-receptor antagonist, in acute heart failure. N Engl J Med. 2010;363(15):1419-28.
- 33. Teerlink JR, Iragui VJ, Mohr JP, Carson PE, Hauptman PJ, Lovett DH, et al. The safety of an adenosine A(1)-receptor antagonist, rolofylline, in patients with acute heart failure and renal impairment: findings from PROTECT. Drug Saf. 2012;35(3):233-44.
- 34. Joo JD, Kim M, Horst P, Kim J, D'Agati VD, Emala CW, Sr., et al. Acute and delayed renal protection against renal ischemia and reperfusion injury with A1 adenosine receptors. Am J Physiol Renal Physiol. 2007;293(6):F1847-57.
- 35. Capurso C, Capurso A. From excess adiposity to insulin resistance: the role of free fatty acids. Vascular pharmacology. 2012;57(2-4):91-7.
- 36. Djousse L, Benkeser D, Arnold A, Kizer JR, Zieman SJ, Lemaitre RN, et al. Plasma free fatty acids and risk of heart failure: the Cardiovascular Health Study. Circulation Heart failure. 2013;6(5):964-9.
- 37. Staehr PM, Dhalla AK, Zack J, Wang X, Ho YL, Bingham J, et al. Reduction of free fatty acids, safety, and pharmacokinetics of oral GS-9667, an A(1) adenosine receptor partial agonist. J Clin Pharmacol. 2013;53(4):385-92.
- 38. Razeghi P, Young ME, Alcorn JL, Moravec CS, Frazier OH, Taegtmeyer H. Metabolic gene expression in fetal and failing human heart. Circulation. 2001;104(24):2923-31.
- 39. Sack MN, Kelly DP. The energy substrate switch during development of heart failure: gene regulatory mechanisms (Review). Int J Mol Med. 1998;1(1):17-24.
- 40. Thum T, Galuppo P, Wolf C, Fiedler J, Kneitz S, van Laake LW, et al. MicroRNAs in the human heart: a clue to fetal gene reprogramming in heart failure. Circulation. 2007;116(3):258-67.

## Integrated Clinical Study Protocol No. BAY 1067197 / 15128



77 FEB 2017 Version: 2.0 

- 41. Albrecht-Kupper BE, Leineweber K, Nell PG. Partial adenosine A1 receptor agonists for cardiovascular therapies. Purinergic signalling. 2012;8(Suppl 1):91-9.
- 42. Sabbah HN, Shimoyama H, Kono T, Gupta RC, Sharov VG, Scicli G, et al. Effects of long-term monotherapy with enalapril, metoprolol, and digoxin on the progression of left ventricular dysfunction and dilation in dogs with reduced ejection fraction. Circulation. 1994;89(6):2852-9.
- 43. Murray AJ, Anderson RE, Watson GC, Radda GK, Clarke K. Uncoupling proteins in human heart. Lancet. 2004;364(9447):1786-8.
- 44. Kelly RP, Ting CT, Yang TM, Liu CP, Maughan WL, Chang MS, et al. Effective arterial elastance as index of arterial vascular load in humans. Circulation. 1992;86(2):513-21.
- 45. The Criteria Committee of the New York Heart Association. Nomenclature and Criteria for Diagnosis of Diseases of the Heart and Great Vessels. 9th ed. Boston, Mass: Little Brown & Co; 1994. p. 253-6.
- 46. Bretz F, Pinheiro JC, Branson M. Combining multiple comparisons and modeling techniques in dose-response studies. Biometrics. 2005;61(3):738-48.
- 47. Carpenter JR, Kenward MG. Missing data in randomized controlled trials a practical guide. Chapter 6.2008.
- 48. Levey AS, Coresh J, Greene T, Stevens LA, Zhang YL, Hendriksen S, et al. Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. Annals of internal medicine. 2006;145(4):247-54.
- 49. Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. The British journal of surgery. 1973;60(8):646-9.




#### 15. Protocol amendments

#### 15.1 Amendment 2

The purpose of Amendment 2 is to implement clarifications after review by regulatory authorities and IRBs and to correct minor errors or omissions.

## 15.1.1 Overview of changes

## 15.1.1.1 Modification 1 – justification of the dose added

Additional wording on the justification of the study drug dose was included.

Affected section: Section 5.3 Justification of the design

## 15.1.1.2 Modification 2 – update in exclusion criteria

- Exclusion criterion related to asthma: a separate criterion for asthma was created to more clearly describe the condition.
- Exclusion criterion related to prohibited therapy was corrected to align with the Investigator Brochure.
- Exclusion criterion related to allergies or hypersensitivities was modified to also exclude patients that are intolerant or hypersensitive to the study treatment.

Affected sections:

- Section 2 Synopsis
- Section 6.2 Exclusion criteria
- Section 8.1.1 Prohibited concomitant medication

## 15.1.1.3 Modification 3 – update to withdrawal section

The withdrawal criterion related to the use of investigational drug other than the study drug was moved from the "*must*" category to the "*may*" category (but recent or concomitant participation in another clinical trial at study entry must still be excluded). Concomitant use of other investigational drugs during the study does not lead to withdrawal from the study. If parallel participation in another study is judged harmful for the patient or there is a possibility of drug-drug interactions that would impact analyses (e.g. PK sampling or ECG), the patient will be withdrawn from the study treatment. However, the patient should preferably still stay in the study for follow-up safety assessments and Week 26 phone call. If the patient is completely withdrawn from the study, no follow-up information can be collected, which will increase the amount of missing data.

Affected section: Section 6.4.1 Withdrawal criteria

## 15.1.1.4 Modification 4 – change in tablet assignment

Tablet combination for patients in 10 mg and 20 mg dose arms was changed as a result of the update on the study drug packaging.

Affected section: Section 7.5 Blinding




## 15.1.1.5 Modification 5 – prohibited medications use – guidance added

Guidance was added for the cases when prohibited medications are taken.

Affected section: Section 8.1.1 Prohibited concomitant medication

# 15.1.1.6 Modification 6 – guidance on concomitant use of BCRP substrates – text added

Information concerning a weak drug-drug interaction with BCRP substrates has been included based on recent availability of phase I data.

Affected section: Section 8.1.2 Permitted therapy

## 15.1.1.7 Modification 7 – updated wording for CEC description

Clinical events for adjudication in Section 13.1 were corrected to be consistent with events defined as secondary efficacy variables in Section 10.3.1.2. "Manual" was replaced by "charter".

Affected section: Section 13.1 Investigator(s) and other study personnel

# 15.1.1.8 Modification 8 – updated statistical calculations for dose-response expressions

Dose-response expressions for the shapes in the candidate sets for change in log-transformed NT-proBNP were updated to align with the SAP

Affected section: Section 10.3.2.2 Analysis of the primary efficacy variables.

### 15.1.1.9 Modification 9 – minor corrections and clarifications

Minor changes were made for better clarity and consistency.

Affected sections:

- Section 2 Synopsis
- Section 3.2 Partial adenosine A1 receptor agonism in heart failure
- Section 6.2 Exclusion criteria
- Section 7.5 Blinding
- Section 9.1 Tabular schedule of evaluations
- Section 9.2 Visit description
- Section 9.4.2 Biomarker investigations
- Section 9.6.3.5 AVIVO monitoring
- Section 10.3.1.3 Other exploratory variables
- Section 11.1 Data recording




## 15.1.2 Changes to the protocol text

All changes are presented in this section by <u>underlining</u> additions and <del>crossing out</del> deletions. Editorial changes and correction of typos are not highlighted in this section.

## 15.1.2.1 Section 2 Synopsis

This section was changed as a result of Modifications 2 and 9.

The same changes were made in the exclusion criteria of the synopsis as the ones detailed in Section 15.1.2.4.

## 15.1.2.2 Section 3.2 Partial adenosine A1 receptor agonism in heart failure

This section was changed as a result of Modification 9.

Old text:

Inhibition of the A1R may also inhibit norepinephrine release from cardiac presynaptic nerves (28, 29).

New text:

Activation of the A1R may also inhibit norepinephrine release from cardiac presynaptic nerves (28, 29).

## 15.1.2.3 Section 5.3 Justification of the design

This section was changed as a result of Modification 1.

Added text:

Evidence of A1R target engagement could already be achieved in different tissues across different clinical trials with 20 mg neladenoson bialanate. The dose range around 20 mg (5, 10, 30 and 40 mg) is to ensure different data points to feed the MCP-Mod predefined models and potential unforeseen variances. The doses studied will ensure a strong dose recommendation moving forward into phase III.

#### 15.1.2.4 Section 6.2 Exclusion criteria

This section was changed as a result of Modifications 2 and 9.

Added text:

- 7. Sustained  $^1$  systolic blood pressure  $\leq$  90 mmHg and / or signs and symptoms of hypotension prior to randomization
- 8. Sustained  $\frac{1}{2}$  systolic blood pressure  $\geq 160$  mmHg
- 9. Sustained <sup>1</sup>-bradycardia with heart rate < 50 beats/minute or tachycardia with heart rate At two consecutive visits.




#### Old text:

- 14. Severe pulmonary disease with any of the following:
  - o Requirement of continuous (home) oxygen or
  - $\circ$  History of chronic obstructive pulmonary disease  $\geq$  GOLD III or
  - Asthma bronchiale

#### *New text:*

- 14. Severe pulmonary disease with any of the following:
  - o Requirement of continuous (home) oxygen or
  - o History of chronic obstructive pulmonary disease ≥ GOLD III or
  - Use of systemic corticosteroids
- 15. Asthma bronchiale with any of the following:
  - o Symptoms not well-controlled within the past 6 months or
  - o Ever intubated or in an intensive care unit for asthma

#### Old text:

- 19. Concomitant use of any of the following therapy that cannot be discontinued:
  - Potent-CYP3A4 inhibitors or inducers or strong CYP2C8 inhibitors (Of note: grapefruit is a strong CYP3A4 inhibitor.)
  - o Theophylline
  - o Drugs that are mainly metabolized by UGT1A1 (irinotecan)

#### *New text:*

- 20. Concomitant use of any of the following therapy that cannot be discontinued:
  - Moderate or strong CYP3A4 inhibitors (Of note: grapefruit is also a strong CYP3A4 inhibitor.)
  - o CYP3A4 inducers
  - o Strong CYP2C8 inhibitors (Of note: clopidogrel is a strong CYP2C8 inhibitor)
  - o Theophylline
  - o Drugs <u>having significant pre-systemic clearance via UGT1A1 in the intestine</u>

#### Old text:

21. Heavy alcohol consumption or the use of illicit drugs that, in the opinion of the investigator, may interfere with the patient's safety and / or compliance

#### New text:

22. Known current heavy alcohol consumption or the use of illicit drugs that, in the opinion of the investigator, may interfere with the patient's safety and / or compliance




Old text:

22. Use of other investigational drugs. Previous (within 30 days or 5 half-lives of the investigational drug, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s)

*New text:* 

<u>23</u>. Previous (within 30 days or 5 half-lives of the investigational drug, whichever is longer) or concomitant participation in another clinical study with investigational medicinal product(s) or device(s)

Old text:

26. Known allergies or hypersensitivities to adhesives or hydrogel

New text:

<u>27</u>. Known allergies, <u>intolerance</u> or hypersensitivities to <u>the study treatment (active substance or excipients)</u>, adhesives or hydrogel

## 15.1.2.5 Section 6.4.1 Withdrawal criteria

This section was changed as a result of Modification 3.

Old text:

Patients *must* be withdrawn from the study if any of the following occurs:

- [...]
- If any investigational drug other than the study drug is used during the study period.

*New text:* 

Patients *may* be withdrawn from the study if any of the following occurs:

- [...]
- If any investigational drug other than the study drug is used during the study period.

## **15.1.2.6 Section 7.5 Blinding**

This section was changed as a result of Modifications 4 and 9.

*Old text:* 

Table 7–3: Assignment of tablets to dose groups

| Treatment arm/<br>Formulation | 5 mg | 10 mg | 20 mg | 30 mg | 40 mg | Placebo |
|---|---|---|---|---|---|---|
| 5 mg | 1 | <del>2</del> | 0 | 0 | 0 | 0 |
| 10 mg | 0 | 0 | <del>2</del> | 1 | 0 | 0 |
| 20 mg | 0 | 0 | 0 | 1 | 2 | 0 |
| Placebo | 1 | 0 | 0 | 0 | 0 | 2 |
| Total tablets/day | 2 | 2 | 2 | 2 | 2 | 2 |




*New text:* 

Table 7-3: Assignment of tablets to dose groups

| Treatment arm/<br>Formulation | 5 mg | 10 mg | 20 mg | 30 mg | 40 mg | Placebo |
|---|---|---|---|---|---|---|
| 5 mg | 1 | 0 | 0 | 0 | 0 | 0 |
| 10 mg | 0 | <u>1</u> | <u>0</u> | 1 | 0 | 0 |
| 20 mg | 0 | 0 | <u>1</u> | 1 | 2 | 0 |
| Placebo | 1 | <u>1</u> | <u>1</u> | 0 | 0 | 2 |
| Total tablets/day | 2 | 2 | 2 | 2 | 2 | 2 |

Added text:

The following parties will be unblinded: sponsor's IxRS and Medication Manager, Clinical Supply Manager and Clinical Pharmacometrics analyst (who will be provided with a randomization list for selected bioanalyses of the active metabolite BAY 84-3174 in plasma), the drug supply's Project Manager, and the DMC.

For all other <u>sponsor's</u> study personnel, the Steering Committee and the Clinical Events Committee (CEC) the blinding will be strictly kept.

### 15.1.2.7 Section 8.1.1 Prohibited concomitant medication

This section was changed as a result of Modifications 2 and 5.

The same changes were made to the list of excluded medications as described in Section 15.1.2.4. In addition, the following text was added:

A list of prohibited medications will be provided to the investigators.

If a prohibited concomitant medication (e.g. moderate / strong CYP3A4 inhibitor) is used during the study conduct, the study drug should be interrupted immediately and restarted as soon as possible, when the prohibited medication has been stopped. Prior to re-starting the study drug, a washout period of at least two days after discontinuation of the prohibited medication should be adhered to.

## 15.1.2.8 Section 8.1.2 Permitted therapy

This section was changed as a result of Modification 6.

Added text:

Neladenoson bialanate is a weak Breast Cancer Resistance Protein (BCRP) inhibitor. The risk of clinically relevant drug—drug interactions at doses up to 40 mg BAY 1067197 due to inhibition of BCRP is regarded as low, but cannot be excluded (BCRP substrates are atorvastatin, simvastatin, rosuvastatin, fluvastatin, methotrexate, etc.; a list of BCRP substrates will be made available to the investigators).

If neladenoson bialanate is given concomitantly with other drugs that may increase the exposure of BCRP substrates, the respective drug labels should be consulted.




## 15.1.2.9 Section 9.1 Tabular schedule of evaluations

This section was changed as a result of Modification 9.

Old text ("dots" were replaced by "pre-dose"):

| Week Day and allowed deviations | <b>-1</b><br>-7 | <b>W0</b><br>0+2 |
|---------------------------------|-----------------|------------------|
| Blood sample for safety | | • |
| Blood sample for biomarkers | | • |
| Urine sample for biomarkers | | • |

#### New text:

| Week Day and allowed deviations | <b>-1</b><br>-7 | <b>W0</b><br>0+2 |
|---------------------------------|-----------------|---------------------|
| Blood sample for safety | | <u>pre-</u><br>dose |
| Blood sample for biomarkers | | <u>pre-</u><br>dose |
| Urine sample for biomarkers | | <u>pre-</u><br>dose |

#### *Old text:*

g [...] If a patient does not take the study drug before the visit, he / she can take it at the start of the visit, in which case PK sampling will occur 2 and 4 hours after the study drug intake.

New text:

g [...] If a patient does not take the study drug before the visit, he / she can take it at the start of the visit, in which case PK sampling will occur <u>as described above</u>.

## **15.1.2.10** Section 9.2 Visit description

This section was changed as a result of Modification 9.

*The following sentence was added to Visit 4 (Week 4) and Visit 5 (Week 8):* 

<u>Ideally</u>, the study personnel should contact the subject prior to Visit 4/Visit 5 to remind them not to take the study drug as usual in the morning at home.

## 15.1.2.11 Section 9.4.2 Biomarker investigations

This section was changed as a result of Modification 9.

Deleted text:

Mandatory (sampled at all time points):

- High sensitivity troponin T (hs-TNT) (baseline disease status & safety)
- Cystatin C (baseline disease status, safety & efficacy)




## **15.1.2.12 Section 9.6.3.5 AVIVO monitoring**

This section was changed as a result of Modification 9.

Old text:

Apart from safety assessments, also the patient's everyday physical activity (frequency, duration, intensity) will be tracked.

*New text:* 

Apart from safety assessments, also the patient's everyday physical activity (<u>e.g.</u> duration, intensity) will be tracked.

## 15.1.2.13 Section 10.3.1.3 Other exploratory variables

This section was changed as a result of Modification 9.

Old text:

• Activity (frequency, duration, intensity) reported values and absolute change from baseline at 20 weeks

*New text:* 

• Activity (duration, intensity) reported values and absolute change from baseline at 20 weeks

## 15.1.2.14 Section 10.3.2.2 Analysis of the primary efficacy variables

This section was changed as a result of Modification 8.

*Old text:* 

Table 10-1: Dose-response shapes used in the candidate set

| Model | Response as function of dose d | |
|---|---|---|
| | LVEF | NT-proBNP |
| Linear | 2 + 0.075 <i>d</i> | -0.105 - 0.005425d |
| Sigmoidal E <sub>max</sub> 1 | $2 + 3.007689d^4 / (9^4 + d^4)$ | $-0.105 - 0.21756d^4 / (9^4 + d^4)$ |
| Sigmoidal E <sub>max</sub> 2 | $2 + 3.375d^3 / (20^3 + d^3)$ | $-0.105 - 0.24413d^3 / (20^3 + d^3)$ |
| E <sub>max</sub> | 2 + 3.09375d / (1.25 + d) | -0.105 - 0.22378d / (1.25 + d) |
| Quadratic | $2 + 0.2d - 0.00333d^2$ | $-0.105 - 0.01447d + 0.00241d^2$ |

New text:

Table 10–1: Dose-response shapes used in the candidate set

| Model | Response as function of dose d | |
|---|---|---|
| | LVEF NT-proBNP | |
| Linear | 2 + 0.075 <i>d</i> | <u>-0.105 - 0.0063<i>d</i></u> |
| Sigmoidal E <sub>max</sub> 1 | $2 + 3.007689d^4 / (9^4 + d^4)$ | $-0.105 - 0.2526d^4 / (9^4 + d^4)$ |
| Sigmoidal E <sub>max</sub> 2 | $2 + 3.375d^3 / (20^3 + d^3)$ | $-0.105 - 0.2835d^3 / (20^3 + d^3)$ |
| E <sub>max</sub> | 2 + 3.09375d / (1.25 + d) | -0.105 - 0.2599d / (1.25 + d) |
| Quadratic | $2 + 0.2d - 0.00333d^2$ | $\underline{-0.105 - 0.0168d + 0.00028d^2}$ |




## 15.1.2.15 Section 11.1 Data recording

This section was changed as a result of Modification 9.

Added text:

Patient data necessary for analysis and reporting will be entered / transmitted into a validated database or data system (e.g. TOSCA; SAS).

## 15.1.2.16 Section 13.1 Investigator(s) and other study personnel

This section was changed as a result of Modification 7.

Old text:

#### **Clinical Events Committee**

Blinded adjudication of all hospitalizations and deaths will be performed by a central CEC as described in the CEC manual. Data entry procedures and documentation necessary for case adjudication will also be described in the CEC manual.

New text:

#### **Clinical Events Committee**

Blinded adjudication of all hospitalizations, <u>urgent visits for HF</u> and deaths will be performed by a central CEC as described in the CEC <u>charter</u>. Data entry procedures and documentation necessary for case adjudication will also be described in the CEC charter.




# 16. Appendices

# 16.1 Calculating glomerular filtration rate

In accordance with established nephrology practice and guidelines, renal function at baseline and throughout the study will be assessed by means of the estimated glomerular filtration rate (eGFR), calculated using the Modification of Diet in Renal Disease (MDRD) study abbreviated formula.

## Isotope dilution mass spectroscopy (IDMS)-traceable MDRD Study Equation:

Conventional units (serum creatinine level is measured in mg/dL)

GFR (mL/min/1.73 m<sup>2</sup>) = 175 x (serum creatinine)<sup>-1.154</sup> x (Age)<sup>-0.203</sup> x (0.742 if female) x (1.212 if African American)

GFR can be estimated using the calculator provided in the following link: http://www.kidney.org/professionals/kdoqi/gfr calculator

For further information on assessing renal function using GFR estimates, see reference (48).

## 16.2 Calculating the Child-Pugh score

The severity of liver disease (Table 16–1) will determine the Child-Pugh score (Table 16–2).

Table 16-1: Grading of severity of liver disease

| Factor | +1 | +2 | +3 |
|--------------------------------|-------|--------------|-------------------|
| Bilirubin (mg/dL) | < 2 | 2 – 3 | > 3 |
| Albumin (g/dL) | > 3.5 | 2.8 - 3.5 | < 2.8 |
| International Normalized Ratio | < 1.7 | 1.7 – 2.3 | > 2.3 |
| Ascites | None | Mild | Moderate / Severe |
| Encephalopathy | None | Grade I - II | Grade III – IV |

Source: adapted from (49)

Table 16-2: Classification using the added score from Table 16-1

| Child-Pugh Class | Α | В | С |
|------------------|-------|-------|---------|
| Points | 5 – 6 | 7 – 9 | 10 – 15 |

Source: adapted from (49)